CLINICAL TRIAL: NCT02907619
Title: A MULTICENTER, OPEN-LABEL EXTENSION STUDY TO EVALUATE THE LONG TERM SAFETY OF PF-06252616 IN BOYS WITH DUCHENNE MUSCULAR DYSTROPHY
Brief Title: An Open-label Extension Study To Evaluate Safety Of PF-06252616 In Boys With Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination Date: 30Aug2018; Reason for termination: Lack of Efficacy
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: B5161004; 2016-001615-21 (EudraCT Number)
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne muscular dystrophy, myostatin, open-label
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — domagrozumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06252616 (Experimental): Either 5mg/kg, 20mg/kg or 40mg/kg will be assigned to a subject based on their maximum tolerated dose from B5161002
  Interventions: Biological: PF-06252616

INTERVENTIONS:
Biological: PF-06252616 — Either 5mg/kg, 20mg/kg or 40mg/kg will be assigned to a subject based on their maximum tolerated dose from B5161002

SUMMARY:
This study is an open-label extension to protocol B5161002 and will provide an assessment of the long term safety, efficacy, pharmacodynamics and pharmacokinetics of intravenous dosing of PF 06252616 in boys with Duchenne muscular dystrophy. Approximately 105 eligible subjects will be assigned to receive a monthly individualized maximum tolerated dose based on their tolerability profile/data from B5161002. This study will not contain a placebo comparator. Subjects will undergo safety evaluations (Laboratory, cardiac monitoring, physical exams, x-ray, MRI), functional capacity evaluations (4 stair climb, range of motion, strength testing, Northstar Ambulatory Assessment, upper limb functional testing, six minute walk test and pulmonary function tests) and pharmacokinetic testing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Duchenne muscular dystrophy who enrolled and completed study B5161002.
2. Signed and dated informed consent document (ICD) indicating that the subject's parent or legal guardian/caregiver has been informed of all pertinent aspects of the study.
3. Subjects and their legal guardians/caregivers who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
4. Subject have;

   1. Adequate hepatic function on screening laboratory assessments
   2. GLDH less than 20 units/liter (2 x upper limit of normal [ULN])
   3. Iron content estimate on the liver MRI within the normal range.

Exclusion Criteria:

1. Unwilling or unable (eg, metal implants) to undergo examination with closed MRI.
2. All male subjects who are able to father children and are sexually active and at risk for impregnating a female partner, who are unwilling or unable to use a highly effective method of contraception. In addition, all sexually active male subjects who are unwilling or unable to prevent potential transfer of and exposure to drug through semen to their partners by using a condom consistently and correctly. .
3. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are related to Pfizer employees directly involved in the conduct of the study.
4. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation.
5. Participation in other studies involving investigational drug(s), with the exception of B5161002.
6. History of allergic or anaphylactic reaction to a therapeutic or diagnostic protein or additives of this investigational product.

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 59 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- United States (26):
  - David Geffen School of Medicine at UCLA/UCLA Neurology, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Pharmacy, Los Angeles, California
  - UCLA (David Geffen School of Medicine), Department of Orthopedic Surgery, Los Angeles, California
  - UCLA Clinical & Translational Research Center, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - University of Iowa ICTS, Clinical Research Unit, Iowa City, Iowa
  - Kennedy Krieger Institute Out-patient Center, Baltimore, Maryland
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Investigational Drug Service, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - (For Drug deliveries) IDS Pharmacy, Minneapolis, Minnesota
  - St. Louis Childrens's Hospital, St Louis, Missouri
  - Duke University Medical Center, Lenox Baker Children's Hospital, Durham, North Carolina
  - Duke University, Investigational Drug Pharmacy, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Center for Clinical and Translational Sciences, Salt Lake City, Utah
  - Utah Center for Advanced Imaging and Research (UCAIR), Salt Lake City, Utah
  - Investigational Drug Services, Salt Lake City, Utah
  - Utah Program for Inherited Neuromuscular Disorder, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - UBC Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Children's Hospital- London Health Sciences Centre, London, Ontario
  - Centre de Readaptation Marie Enfant (CRME), Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
- Italy (9):
  - UOC Farmacia - Istituto Gianna Gaslini,, Genova
  - UOC Medicina Fisica Riabilitativa - Istituto G. Gaslini, Genova
  - UOC Neurologia Pediatrica e Malattie Muscolari Istituto Gianna Gaslini, Genova
  - UOC Radiologia - Istituto Gianna Gaslini,, Genova
  - UOS Dipartimentale Endocrinologia Clinica Sperimentale - Ist., Genova
  - Dipartimento Pediatrico Universitario-Ospedaliero Endocrinologia, Rome
  - Farmacia Ospedaliera, IRCCS Ospedale Pediatrico Bambino Gesu, Rome
  - IRCCS Ospedale Pediatrico Bambino Gesu - Centro Trials, Rome
  - U.O. Malattie Neuromuscolari e Neurodegenerative, IRCCS Ospedale Pediatrico Bambino Gesu, Rome
- Japan (2):
  - Hyogo college of medicine hospital, Nishinomiya-shi, Hyōgo
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
- United Kingdom (5):
  - Dubowitz Neuromuscular Centre, Institute of Child Health, London
  - Great Ormond Street Hospital, London
  - Institute of Genetic Medicine,Muscle Team, Newcastle upon Tyne
  - Clinical Research Facility, Newcastle upon Tyne
  - Royal Victoria Infirmary Research Pharmacy, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wagner KR, Abdel-Hamid HZ, Mah JK, Campbell C, Guglieri M, Muntoni F, Takeshima Y, McDonald CM, Kostera-Pruszczyk A, Karachunski P, Butterfield RJ, Mercuri E, Fiorillo C, Bertini ES, Tian C, Statland J, Sadosky AB, Purohit VS, Sherlock SP, Palmer JP, Binks M, Charnas L, Marraffino S, Wong BL. Randomized phase 2 trial and open-label extension of domagrozumab in Duchenne muscular dystrophy. Neuromuscul Disord. 2020 Jun;30(6):492-502. doi: 10.1016/j.nmd.2020.05.002. Epub 2020 May 19. PMID 32522498
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B5161004

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study B5161004 was an open-label extension (OLE) to study B5161002. The parent study B5161002 was a Phase 2, randomized, 2-period, blinded, placebo controlled study to evaluate the safety, efficacy, PK and PD of domagrozumab administered to ambulatory boys diagnosed with DMD.
Groups:
- Sequence 1: In study B5161002 (parent study) participants randomized to Sequence group 1 received domagrozumab (PF-06252616) in a dose escalating fashion (5, 20 and 40 mg/kg) in Period 1. At each dose level, domagrozumab was administered over 2 hours by intravenous (IV) infusion every 4 weeks for a total of 16 weeks. In Period 2, participants received domagrozumab every 4 weeks for a total of 48 weeks at 40 mg/kg, the maximum tolerated dose identified in Period 1. There was no pause between Period 1 and Period 2 (48 weeks each). In study B5161004 (OLE) participants received domagrozumab 40 mg/kg every 4 weeks until early termination of this study. The OLE study reports participants within the treatment assignment they received in the parent study.
- Sequence 2: In study B5161002 (parent study) participants randomized to Sequence group 2 received domagrozumab (PF-06252616) in a dose escalating fashion (5, 20 and 40 mg/kg) in Period 1. At each dose level, domagrozumab was administered over 2 hours by IV infusion every 4 weeks for a total of 16 weeks. In Period 2, participants received placebo. There was no pause between Period 1 and Period 2 (48 weeks each). In study B5161004 (OLE) participants received domagrozumab 40 mg/kg (the maximum tolerated dose from B5161002) every 4 weeks until early termination of this study. The OLE study reports participants within the treatment assignment they received in the parent study.
- Sequence 3: In study B5161002 (parent study) participants randomized to Sequence group 3 received placebo in Period 1 (48 weeks). In Period 2, participants received domagrozumab (PF-06252616) in a dose escalating fashion (5, 20 and 40 mg/kg). At each dose level, domagrozumab was administered over 2 hours by IV infusion every 4 weeks for a total of 16 weeks. There was no pause between Period 1 and Period 2 (48 weeks each). In study B5161004 (OLE) participants received domagrozumab 40 mg/kg (the maximum tolerated dose from B5161002) every 4 weeks until early termination of this study. The OLE study reports participants within the treatment assignment they received in the parent study.
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Started | 19 | 20 | 20
Received Treatment | 19 | 20 | 20
Completed | 0 | 0 | 0
Not Completed | 19 | 20 | 20
Not completed — Study terminated by sponsor | 18 | 18 | 19
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment in this study B5161004.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 20 | 20 | 59
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.0) | 10.2 (0.9) | 10.4 (1.1) | 9.9 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 19 | 20 | 20 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18 | 17 | 18 | 53
  Asian | 1 | 2 | 2 | 5
  Other | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Reduced or Temporary Discontinuation Due to AEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment or usage. Treatment-related AEs were determined by the investigator. The number of participants with dose reduced or temporary discontinuation due to both all-causality and treatment-related AEs are presented below.
Time Frame: 2 Years
Population: The analysis population included all participants who had received at least 1 dose of study medication in current study B5161004.
Measure: Count of Participants; unit: Participants
Groups:
- Total: Sum of all participants in the study B5161004
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Due to All-causality AEs | 0 | 0 | 0 | 0
  Due to Treatment-related AEs | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Severe Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment or usage. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment. Severe TEAEs were TEAEs that interfered significantly with participants' usual function. Treatment-related TEAEs were determined by the investigator. The number of participants with severe all-causality and treatment-related TEAEs are presented below.
Time Frame: 2 Years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  All-Causality TEAEs | 3 | 0 | 1 | 4
  Treatment-Related TEAEs | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Who Discontinued From the Study Due to TEAEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a product; the event did not need to have a causal relationship with the treatment or usage. TEAEs were AEs occurred following the start of treatment or AEs increasing in severity during treatment. Treatment-related TEAEs were determined by the investigator. The number of participants who discontinued from the study due to both all-causality and treatment-related TEAEs are presented below.
Time Frame: 2 Years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Due to All-causality AEs | 0 | 0 | 1 | 1
  Due to Treatment-related AEs | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to B5161004 Baseline Abnormality) - Hematology
Description: Hematology evaluation included: hemoglobin, hematocrit, red blood cell (RBC) count, platelets, RBC morphology, white blood cell (WBC) count, absolute lymphocytes, absolute atypical lymphocytes, absolute total neutrophils, absolute total neutrophils count, absolute band cells, absolute basophils, absolute eosinophils and absolute monocytes.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004.
  (ULN=Upper Limit of Normal; LLN=Lower Limit of Normal).
Time Frame: 2 Years
Population: Analysis population included all participants who had received at least 1 dose of study medication in current study B5161004. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Hemoglobin <0.8 × LLN | 0 | 0 | 0 | 0
  Hematocrit <0.8 × LLN | 0 | 0 | 0 | 0
  RBC count <0.8 × LLN | 0 | 0 | 0 | 0
  Platelets <0.5 × LLN | 0 | 0 | 0 | 0
  Platelets >1.75 × ULN | 0 | 0 | 0 | 0
  RBC Morphology >0 | 0 | 1 | 0 | 1
  WBC count <0.6 × LLN | 0 | 0 | 0 | 0
  WBC count >1.5 × ULN | 0 | 0 | 0 | 0
  Absolute Lymphocytes <0.8 × LLN | 0 | 0 | 0 | 0
  Absolute lymphocytes >1.2 × ULN | 0 | 0 | 0 | 0
  Absolute atypical lymphocytes >0: number analyzed (Participants) | 1 | 0 | 0 | 1
  Absolute atypical lymphocytes >0 | 1 |  |  | 1
  Absolute total neutrophils <0.8 × LLN | 0 | 0 | 0 | 0
  Absolute total neutrophils >1.2 × ULN | 3 | 1 | 2 | 6
  Absolute total neutrophil count <1.35 × 10^3/mcL | 0 | 0 | 0 | 0
  Absolute total neutrophil count >8.15 × 10^3/mcL | 6 | 1 | 5 | 12
  Absolute band cells >0.27 × 10^3/mcL: number analyzed (Participants) | 1 | 0 | 0 | 1
  Absolute band cells >0.27 × 10^3/mcL | 0 |  |  | 0
  Absolute basophils >1.2 × ULN | 0 | 0 | 0 | 0
  Absolute eosinophils >1.2 × ULN | 1 | 0 | 1 | 2
  Absolute monocytes >1.2 × ULN | 1 | 0 | 1 | 2

5. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to B5161004 Baseline Abnormality) - Coagulation
Description: Coagulation evaluation included activated partial thromboplastin time (aPTT) and prothrombin time (PT).
  (ULN=Upper Limit of Normal). Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004.
Time Frame: 2 Years
Population: Analysis population included all participants who had received at least 1 dose of study medication in current study B5161004.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  aPTT >1.1 x ULN | 0 | 0 | 1 | 1
  PT >1.1 x ULN | 1 | 0 | 1 | 2

6. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to B5161004 Baseline Abnormality) - Liver Function
Description: Liver function evaluation included: total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), alkaline phosphatase, total protein, albumin and glutamate dehydrogenase.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004.
  (LLN=Lower Limit of Normal; ULN=Upper Limit of Normal).
Time Frame: 2 Years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Total Bilirubin >1.5 x ULN | 0 | 0 | 0 | 0
  AST >3.0 x ULN | 16 | 16 | 15 | 47
  ALT >3.0 x ULN | 19 | 18 | 19 | 56
  GGT >3.0 x ULN | 0 | 0 | 0 | 0
  Alkaline Phosphatase >3.0 x ULN | 0 | 0 | 0 | 0
  Total Protein <0.8 x LLN | 0 | 0 | 0 | 0
  Total Protein >1.2 x ULN | 0 | 0 | 0 | 0
  Albumin <0.8 x LLN | 0 | 0 | 0 | 0
  Albumin >1.2 x ULN | 0 | 0 | 0 | 0
  Glutamate Dehydrogenase >1.0 x ULN | 0 | 0 | 1 | 1

7. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to B5161004 Baseline Abnormality) - Renal Function
Description: Renal function evaluation included: blood urea nitrogen (BUN), creatinine and uric acid.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. (ULN=Upper Limit of Normal).
Time Frame: 2 Years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Blood Urea Nitrogen (BUN) >1.3 x ULN | 0 | 0 | 0 | 0
  Creatinine >1.3 x ULN | 0 | 0 | 0 | 0
  Uric Acid >1.2 x ULN | 1 | 0 | 0 | 1

8. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to B5161004 Baseline Abnormality) - Electrolytes
Description: Electrolytes evaluation included: sodium, potassium, chloride, calcium, phosphate and bicarbonate.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004.
  (LLN=Lower Limit of Normal, ULN=Upper Limit of Normal).
Time Frame: 2 Years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Sodium <0.95 x LLN | 0 | 0 | 0 | 0
  Sodium >1.05 x ULN | 0 | 0 | 0 | 0
  Potassium <0.9 x LLN | 0 | 0 | 0 | 0
  Potassium >1.1 x ULN | 1 | 0 | 0 | 1
  Chloride <0.9 x LLN | 0 | 0 | 0 | 0
  Chloride >1.1 x ULN | 0 | 0 | 0 | 0
  Calcium <0.9 x LLN | 0 | 0 | 0 | 0
  Calcium >1.1 x ULN | 0 | 0 | 0 | 0
  Phosphate <0.8 x LLN | 0 | 0 | 0 | 0
  Phosphate >1.2 x ULN | 0 | 0 | 0 | 0
  Bicarbonate (venous) <0.9 x LLN | 0 | 0 | 0 | 0
  Bicarbonate (venous) >1.1 x ULN | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to B5161004 Baseline Abnormality) - Hormones
Description: Hormone evaluations included free thyroxine (T4), thyroid stimulating hormone (TSH), lutenizing hormone (LH), follicle stimulating hormone (FSH), and androstenedione. Numbers of participants with abnormalities of LH, FSH and androstenedione were reported in different age groups.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004.
  (LLN=Lower Limit of Normal, ULN=Upper Limit of Normal).
Time Frame: 2 Years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  T4 (free) <0.8 x LLN: number analyzed (Participants) | 18 | 18 | 17 | 53
  T4 (free) <0.8 x LLN | 0 | 0 | 0 | 0
  T4 (free) >1.2 x ULN: number analyzed (Participants) | 18 | 18 | 17 | 53
  T4 (free) >1.2 x ULN | 0 | 0 | 0 | 0
  TSH <0.8 x LLN: number analyzed (Participants) | 18 | 18 | 17 | 53
  TSH <0.8 x LLN | 0 | 1 | 0 | 1
  TSH >1.2 x ULN: number analyzed (Participants) | 18 | 18 | 17 | 53
  TSH >1.2 x ULN | 0 | 0 | 0 | 0
  LH (7years - <9 years) <0.3mIU/mL: number analyzed (Participants) | 2 | 0 | 0 | 2
  LH (7years - <9 years) <0.3mIU/mL | 0 |  |  | 0
  LH(7years - <9 years) >2.8mIU/mL: number analyzed (Participants) | 2 | 0 | 0 | 2
  LH(7years - <9 years) >2.8mIU/mL | 0 |  |  | 0
  LH (9years - <11 years) <0.3mIU/mL: number analyzed (Participants) | 13 | 5 | 4 | 22
  LH (9years - <11 years) <0.3mIU/mL | 8 | 5 | 3 | 16
  LH (9years - <11 years) >2.8mIU/mL: number analyzed (Participants) | 13 | 5 | 4 | 22
  LH (9years - <11 years) >2.8mIU/mL | 0 | 0 | 0 | 0
  LH (11years - <12 years) <0.3mIU/mL: number analyzed (Participants) | 3 | 6 | 2 | 11
  LH (11years - <12 years) <0.3mIU/mL | 2 | 3 | 2 | 7
  LH (11years - <12 years) >1.8mIU/mL: number analyzed (Participants) | 3 | 6 | 2 | 11
  LH (11years - <12 years) >1.8mIU/mL | 0 | 0 | 0 | 0
  LH(12years - <13 years) <0.3 mIU/mL: number analyzed (Participants) | 1 | 8 | 11 | 20
  LH(12years - <13 years) <0.3 mIU/mL | 0 | 5 | 8 | 13
  LH(12years - <13 years) >4.0mIU/mL: number analyzed (Participants) | 1 | 8 | 11 | 20
  LH(12years - <13 years) >4.0mIU/mL | 0 | 0 | 0 | 0
  LH(13years - <14 years) <0.3mIU/mL: number analyzed (Participants) | 1 | 1 | 1 | 3
  LH(13years - <14 years) <0.3mIU/mL | 1 | 0 | 1 | 2
  LH(13years - <14 years) >6.0mIU/mL: number analyzed (Participants) | 1 | 1 | 1 | 3
  LH(13years - <14 years) >6.0mIU/mL | 0 | 0 | 0 | 0
  FSH(7years - <9 years) >4.10mIU/mL: number analyzed (Participants) | 2 | 0 | 0 | 2
  FSH(7years - <9 years) >4.10mIU/mL | 0 |  |  | 0
  FSH (9years - <11 years) >4.50mIU/mL: number analyzed (Participants) | 13 | 5 | 4 | 22
  FSH (9years - <11 years) >4.50mIU/mL | 0 | 0 | 0 | 0
  FSH (11years - <12 years) <0.40mIU/mL: number analyzed (Participants) | 3 | 6 | 2 | 11
  FSH (11years - <12 years) <0.40mIU/mL | 0 | 0 | 0 | 0
  FSH (11years - <12 years) >8.90mIU/mL: number analyzed (Participants) | 3 | 6 | 2 | 11
  FSH (11years - <12 years) >8.90mIU/mL | 0 | 0 | 0 | 0
  FSH (12years - <13 years) <0.50mIU/mL: number analyzed (Participants) | 1 | 8 | 11 | 20
  FSH (12years - <13 years) <0.50mIU/mL | 0 | 0 | 0 | 0
  FSH (12years - <13 years) >10.50mIU/mL: number analyzed (Participants) | 1 | 8 | 11 | 20
  FSH (12years - <13 years) >10.50mIU/mL | 0 | 0 | 0 | 0
  FSH (13years - <14 years) <0.70mIU/mL: number analyzed (Participants) | 1 | 1 | 1 | 3
  FSH (13years - <14 years) <0.70mIU/mL | 1 | 0 | 1 | 2
  FSH (13 years - <14 years) >10.80mIU/mL: number analyzed (Participants) | 1 | 1 | 1 | 3
  FSH (13 years - <14 years) >10.80mIU/mL | 0 | 0 | 0 | 0
  Androstenedione (7 - <10years) <3 ng/dL: number analyzed (Participants) | 6 | 2 | 4 | 12
  Androstenedione (7 - <10years) <3 ng/dL | 0 | 0 | 2 | 2
  Androstenedione(7 - <10 years) >31 ng/dL: number analyzed (Participants) | 6 | 2 | 4 | 12
  Androstenedione(7 - <10 years) >31 ng/dL | 1 | 1 | 0 | 2
  Androstenedione (10 - <12years) <7 ng/dL: number analyzed (Participants) | 12 | 9 | 2 | 23
  Androstenedione (10 - <12years) <7 ng/dL | 5 | 3 | 1 | 9
  Androstenedione (10-<12years) >41 ng/dL: number analyzed (Participants) | 12 | 9 | 2 | 23
  Androstenedione (10-<12years) >41 ng/dL | 1 | 0 | 0 | 1
  Androstenedione (12 - <14years) <11 ng/dL: number analyzed (Participants) | 1 | 8 | 11 | 20
  Androstenedione (12 - <14years) <11 ng/dL | 1 | 4 | 6 | 11
  Androstenedione (12 - <14years) >64 ng/dL: number analyzed (Participants) | 1 | 8 | 11 | 20
  Androstenedione (12 - <14years) >64 ng/dL | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to B5161004 Baseline Abnormality) - Clinical Chemistry
Description: Clinical chemistry evaluation included glucose, creatine kinase (CK), troponin I, amylase, iron binding capacity, unsaturated iron binding capacity, transferrin saturation, iron and ferritin. Number of participants with iron abnormalities was reported in different age groups.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004.
  (LLN=Lower Limit of Normal, ULN=Upper Limit of Normal).
Time Frame: 2 Years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Glucose <0.6 x LLN | 0 | 0 | 0 | 0
  Glucose >1.5 x ULN | 0 | 0 | 0 | 0
  CK >2.0 x ULN | 19 | 20 | 20 | 59
  Troponin I >3.0 x ULN: number analyzed (Participants) | 19 | 18 | 17 | 54
  Troponin I >3.0 x ULN | 4 | 4 | 1 | 9
  Amylase > 1.5 x ULN | 0 | 0 | 1 | 1
  Iron Binding Capacity <37.6 mcg/dL | 0 | 0 | 0 | 0
  Unsaturated Iron Binding Capacity <130 mcg/dL | 3 | 4 | 3 | 10
  Unsaturated Iron Binding Capacity >375 mcg/dL | 0 | 0 | 0 | 0
  Transferrin Saturation < 20% | 0 | 3 | 2 | 5
  Transferrin Saturation > 50% | 7 | 4 | 6 | 17
  Iron 1Y<=Age<11Y <50: number analyzed (Participants) | 17 | 8 | 6 | 31
  Iron 1Y<=Age<11Y <50 | 0 | 0 | 1 | 1
  Iron 1Y<=Age<11Y >120: number analyzed (Participants) | 17 | 8 | 6 | 31
  Iron 1Y<=Age<11Y >120 | 12 | 2 | 2 | 16
  Iron 11Y<=Age<18Y <50: number analyzed (Participants) | 4 | 15 | 15 | 34
  Iron 11Y<=Age<18Y <50 | 0 | 3 | 0 | 3
  Iron 11Y<=Age<18Y >170: number analyzed (Participants) | 4 | 15 | 15 | 34
  Iron 11Y<=Age<18Y >170 | 0 | 1 | 1 | 2
  Ferritin <15 ng/mL | 4 | 6 | 5 | 15
  Ferritin >140 ng/mL | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to B5161004 Baseline Abnormality) - Urinalysis
Description: Urinalysis Microscopy included: urine red blood cell (RBC), urine white blood cell (WBC), urine uric acid crystals, urine calcium oxalate crystals, urine amorphous crystals, urine bacteria, urine microscopic exam.
  Urinalysis Dipstick included: urine pH, urine glucose, urine ketones, urine protein, urine blood/hemoglobin, urine nitrite, urine leukocyte esterase.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004.
Time Frame: 2 Years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Microscopy - Urine RBC >=20: number analyzed (Participants) | 2 | 3 | 1 | 6
  Microscopy - Urine RBC >=20 | 0 | 0 | 0 | 0
  Microscopy - Urine WBC >=20: number analyzed (Participants) | 6 | 8 | 6 | 20
  Microscopy - Urine WBC >=20 | 0 | 0 | 0 | 0
  Microscopy-Urine Uric Acid Crystals -Present: number analyzed (Participants) | 1 | 0 | 0 | 1
  Microscopy-Urine Uric Acid Crystals -Present | 1 |  |  | 1
  Microscopy-Urine Calcium Oxalate Crystals -Present: number analyzed (Participants) | 4 | 7 | 4 | 15
  Microscopy-Urine Calcium Oxalate Crystals -Present | 4 | 7 | 4 | 15
  Microscopy-Urine Amorphous Crystals -Present: number analyzed (Participants) | 3 | 3 | 2 | 8
  Microscopy-Urine Amorphous Crystals -Present | 3 | 3 | 2 | 8
  Microscopy - Urine Bacteria >20: number analyzed (Participants) | 1 | 1 | 0 | 2
  Microscopy - Urine Bacteria >20 | 0 | 0 |  | 0
  Microscopy-Urine Microscopic Exam -Positive: number analyzed (Participants) | 9 | 11 | 8 | 28
  Microscopy-Urine Microscopic Exam -Positive | 8 | 11 | 7 | 26
  Dipstick - Urine pH <4.5 | 0 | 0 | 0 | 0
  Dipstick - Urine pH >8 | 0 | 1 | 0 | 1
  Dipstick - urine glucose >=1 | 0 | 0 | 0 | 0
  Dipstick - urine ketones >=1 | 0 | 1 | 1 | 2
  Dipstick - urine protein >=1 | 0 | 0 | 0 | 0
  Dipstick - urine blood/hemoglobin >=1 | 0 | 0 | 0 | 0
  Dipstick - Urine nitrite >=1 | 0 | 0 | 0 | 0
  Dipstick - Urine Leukocyte Esterase >=1 | 0 | 1 | 0 | 1

12. Primary Outcome: Number of Participants With Laboratory Test Abnormalities (Without Regard to B5161004 Baseline Abnormality) - Fecal Blood
Description: Number of participants with blood detected in fecal samples is presented. Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004.
  (ULN=Upper Limit of Normal).
Time Frame: 2 Years
Population: Analysis population included all participants who had received at least 1 dose of study medication in current study B5161004 and who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 17 | 17 | 53
Participants | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Data of Serum Ferritin, Serum Iron and % Transferrin Saturation Meeting Categorical Summarization Criteria - B5161004 Baseline
Description: Participants were asked to fast for at least 8 hours prior to collection of blood to evaluate serum iron, serum ferritin and % transferrin saturation. The unit of iron was mcg/dL; the unit of ferritin was ng/mL; the unit of %transferrin saturation was %.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 37, 49, 61, 73 and 85.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Iron - Baseline: <120 | 13 | 18 | 10 | 41
  Iron - Baseline: 120 - <144 | 3 | 2 | 6 | 11
  Iron - Baseline: 144 - <200 | 3 | 0 | 4 | 7
  Iron - Baseline: >=200 | 0 | 0 | 0 | 0
  Iron - Week 13: <120: number analyzed (Participants) | 15 | 16 | 17 | 48
  Iron - Week 13: <120 | 10 | 15 | 9 | 34
  Iron - Week 13: 120 - <144: number analyzed (Participants) | 15 | 16 | 17 | 48
  Iron - Week 13: 120 - <144 | 3 | 0 | 7 | 10
  Iron - Week 13: 144 - <200: number analyzed (Participants) | 15 | 16 | 17 | 48
  Iron - Week 13: 144 - <200 | 2 | 1 | 1 | 4
  Iron - Week 13: >=200: number analyzed (Participants) | 15 | 16 | 17 | 48
  Iron - Week 13: >=200 | 0 | 0 | 0 | 0
  Iron - Week 25: <120: number analyzed (Participants) | 12 | 12 | 13 | 37
  Iron - Week 25: <120 | 8 | 10 | 8 | 26
  Iron - Week 25: 120 - <144: number analyzed (Participants) | 12 | 12 | 13 | 37
  Iron - Week 25: 120 - <144 | 3 | 0 | 4 | 7
  Iron - Week 25: 144 - <200: number analyzed (Participants) | 12 | 12 | 13 | 37
  Iron - Week 25: 144 - <200 | 1 | 2 | 1 | 4
  Iron - Week 25: >=200: number analyzed (Participants) | 12 | 12 | 13 | 37
  Iron - Week 25: >=200 | 0 | 0 | 0 | 0
  Iron-Week 37: <120: number analyzed (Participants) | 8 | 9 | 12 | 29
  Iron-Week 37: <120 | 5 | 6 | 10 | 21
  Iron-Week 37: 120 - <144: number analyzed (Participants) | 8 | 9 | 12 | 29
  Iron-Week 37: 120 - <144 | 1 | 3 | 2 | 6
  Iron-Week 37: 144 - <200: number analyzed (Participants) | 8 | 9 | 12 | 29
  Iron-Week 37: 144 - <200 | 2 | 0 | 0 | 2
  Iron-Week 37: >=200: number analyzed (Participants) | 8 | 9 | 12 | 29
  Iron-Week 37: >=200 | 0 | 0 | 0 | 0
  Iron-Week 49: <120: number analyzed (Participants) | 7 | 6 | 8 | 21
  Iron-Week 49: <120 | 6 | 3 | 6 | 15
  Iron-Week 49: 120 - <144: number analyzed (Participants) | 7 | 6 | 8 | 21
  Iron-Week 49: 120 - <144 | 1 | 0 | 1 | 2
  Iron-Week 49: 144 - <200: number analyzed (Participants) | 7 | 6 | 8 | 21
  Iron-Week 49: 144 - <200 | 0 | 3 | 1 | 4
  Iron-Week 49: >=200: number analyzed (Participants) | 7 | 6 | 8 | 21
  Iron-Week 49: >=200 | 0 | 0 | 0 | 0
  Iron-Week 61: <120: number analyzed (Participants) | 3 | 4 | 3 | 10
  Iron-Week 61: <120 | 1 | 2 | 2 | 5
  Iron-Week 61: 120 - <144: number analyzed (Participants) | 3 | 4 | 3 | 10
  Iron-Week 61: 120 - <144 | 1 | 1 | 1 | 3
  Iron-Week 61: 144 - <200: number analyzed (Participants) | 3 | 4 | 3 | 10
  Iron-Week 61: 144 - <200 | 1 | 1 | 0 | 2
  Iron-Week 61: >=200: number analyzed (Participants) | 3 | 4 | 3 | 10
  Iron-Week 61: >=200 | 0 | 0 | 0 | 0
  Iron-Week 73: <120: number analyzed (Participants) | 2 | 2 | 2 | 6
  Iron-Week 73: <120 | 1 | 1 | 2 | 4
  Iron-Week 73: 120 - <144: number analyzed (Participants) | 2 | 2 | 2 | 6
  Iron-Week 73: 120 - <144 | 1 | 0 | 0 | 1
  Iron-Week 73: 144 - <200: number analyzed (Participants) | 2 | 2 | 2 | 6
  Iron-Week 73: 144 - <200 | 0 | 1 | 0 | 1
  Iron-Week 73: >=200: number analyzed (Participants) | 2 | 2 | 2 | 6
  Iron-Week 73: >=200 | 0 | 0 | 0 | 0
  Iron-Week 85: <120: number analyzed (Participants) | 0 | 1 | 1 | 2
  Iron-Week 85: <120 | 0 | 1 | 1 | 2
  Iron-Week 85: 120 - <144: number analyzed (Participants) | 0 | 1 | 1 | 2
  Iron-Week 85: 120 - <144 | 0 | 0 | 0 | 0
  Iron-Week 85: 144 - <200: number analyzed (Participants) | 0 | 1 | 1 | 2
  Iron-Week 85: 144 - <200 | 0 | 0 | 0 | 0
  Iron-Week 85: >=200: number analyzed (Participants) | 0 | 1 | 1 | 2
  Iron-Week 85: >=200 | 0 | 0 | 0 | 0
  Ferritin-Baseline: <140 | 19 | 20 | 20 | 59
  Ferritin-Baseline: >=140 | 0 | 0 | 0 | 0
  Ferritin-Week 13: <140: number analyzed (Participants) | 14 | 17 | 16 | 47
  Ferritin-Week 13: <140 | 14 | 17 | 16 | 47
  Ferritin-Week 13: >=140: number analyzed (Participants) | 14 | 17 | 16 | 47
  Ferritin-Week 13: >=140 | 0 | 0 | 0 | 0
  Ferritin-Week 25: <140: number analyzed (Participants) | 12 | 12 | 13 | 37
  Ferritin-Week 25: <140 | 12 | 12 | 13 | 37
  Ferritin-Week 25: >=140: number analyzed (Participants) | 12 | 12 | 13 | 37
  Ferritin-Week 25: >=140 | 0 | 0 | 0 | 0
  Ferritin-Week 37: <140: number analyzed (Participants) | 7 | 9 | 12 | 28
  Ferritin-Week 37: <140 | 7 | 9 | 12 | 28
  Ferritin-Week 37: >=140: number analyzed (Participants) | 7 | 9 | 12 | 28
  Ferritin-Week 37: >=140 | 0 | 0 | 0 | 0
  Ferritin-Week 49: <140: number analyzed (Participants) | 7 | 6 | 8 | 21
  Ferritin-Week 49: <140 | 7 | 6 | 8 | 21
  Ferritin-Week 49: >=140: number analyzed (Participants) | 7 | 6 | 8 | 21
  Ferritin-Week 49: >=140 | 0 | 0 | 0 | 0
  Ferritin-Week 61: <140: number analyzed (Participants) | 2 | 4 | 3 | 9
  Ferritin-Week 61: <140 | 2 | 4 | 3 | 9
  Ferritin-Week 61: >=140: number analyzed (Participants) | 2 | 4 | 3 | 9
  Ferritin-Week 61: >=140 | 0 | 0 | 0 | 0
  Ferritin-Week 73: <140: number analyzed (Participants) | 2 | 2 | 2 | 6
  Ferritin-Week 73: <140 | 2 | 2 | 2 | 6
  Ferritin-Week 73: >=140: number analyzed (Participants) | 2 | 2 | 2 | 6
  Ferritin-Week 73: >=140 | 0 | 0 | 0 | 0
  Ferritin-Week 85: <140: number analyzed (Participants) | 0 | 1 | 1 | 2
  Ferritin-Week 85: <140 | 0 | 1 | 1 | 2
  Ferritin-Week 85: >=140: number analyzed (Participants) | 0 | 1 | 1 | 2
  Ferritin-Week 85: >=140 | 0 | 0 | 0 | 0
  %Transferrin Saturation - Baseline: <45: number analyzed (Participants) | 18 | 20 | 20 | 58
  %Transferrin Saturation - Baseline: <45 | 15 | 20 | 18 | 53
  %Transferrin Saturation Baseline: 45 - <50: number analyzed (Participants) | 18 | 20 | 20 | 58
  %Transferrin Saturation Baseline: 45 - <50 | 3 | 0 | 1 | 4
  %Transferrin Saturation Baseline: 50 - <69: number analyzed (Participants) | 18 | 20 | 20 | 58
  %Transferrin Saturation Baseline: 50 - <69 | 0 | 0 | 1 | 1
  %Transferrin Saturation Baseline: >=69: number analyzed (Participants) | 18 | 20 | 20 | 58
  %Transferrin Saturation Baseline: >=69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 13: <45: number analyzed (Participants) | 15 | 16 | 16 | 47
  %Transferrin Saturation Week 13: <45 | 12 | 15 | 13 | 40
  %Transferrin Saturation Week 13: 45 - <50: number analyzed (Participants) | 15 | 16 | 16 | 47
  %Transferrin Saturation Week 13: 45 - <50 | 1 | 0 | 1 | 2
  %Transferrin Saturation Week 13: 50 - <69: number analyzed (Participants) | 15 | 16 | 16 | 47
  %Transferrin Saturation Week 13: 50 - <69 | 2 | 1 | 2 | 5
  %Transferrin Saturation Week 13: >=69: number analyzed (Participants) | 15 | 16 | 16 | 47
  %Transferrin Saturation Week 13: >=69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 25: <45: number analyzed (Participants) | 10 | 12 | 13 | 35
  %Transferrin Saturation Week 25: <45 | 9 | 10 | 9 | 28
  %Transferrin Saturation Week 25: 45 - <50: number analyzed (Participants) | 10 | 12 | 13 | 35
  %Transferrin Saturation Week 25: 45 - <50 | 0 | 1 | 2 | 3
  %Transferrin Saturation Week 25: 50 - <69: number analyzed (Participants) | 10 | 12 | 13 | 35
  %Transferrin Saturation Week 25: 50 - <69 | 1 | 1 | 2 | 4
  %Transferrin Saturation Week 25: >=69: number analyzed (Participants) | 10 | 12 | 13 | 35
  %Transferrin Saturation Week 25: >=69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 37: <45: number analyzed (Participants) | 6 | 7 | 12 | 25
  %Transferrin Saturation Week 37: <45 | 4 | 6 | 11 | 21
  %Transferrin Saturation Week 37: 45 - <50: number analyzed (Participants) | 6 | 7 | 12 | 25
  %Transferrin Saturation Week 37: 45 - <50 | 1 | 0 | 0 | 1
  %Transferrin Saturation Week 37: 50 - <69: number analyzed (Participants) | 6 | 7 | 12 | 25
  %Transferrin Saturation Week 37: 50 - <69 | 1 | 1 | 1 | 3
  %Transferrin Saturation Week 37: >=69: number analyzed (Participants) | 6 | 7 | 12 | 25
  %Transferrin Saturation Week 37: >=69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 49: <45: number analyzed (Participants) | 7 | 6 | 8 | 21
  %Transferrin Saturation Week 49: <45 | 6 | 4 | 6 | 16
  %Transferrin Saturation Week 49: 45 - <50: number analyzed (Participants) | 7 | 6 | 8 | 21
  %Transferrin Saturation Week 49: 45 - <50 | 0 | 0 | 1 | 1
  %Transferrin Saturation Week 49: 50 - <69: number analyzed (Participants) | 7 | 6 | 8 | 21
  %Transferrin Saturation Week 49: 50 - <69 | 1 | 2 | 1 | 4
  %Transferrin Saturation Week 49: >=69: number analyzed (Participants) | 7 | 6 | 8 | 21
  %Transferrin Saturation Week 49: >=69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 61: <45: number analyzed (Participants) | 1 | 3 | 3 | 7
  %Transferrin Saturation Week 61: <45 | 1 | 2 | 3 | 6
  %Transferrin Saturation Week 61: 45 - <50: number analyzed (Participants) | 1 | 3 | 3 | 7
  %Transferrin Saturation Week 61: 45 - <50 | 0 | 1 | 0 | 1
  %Transferrin Saturation Week 61: 50 - <69: number analyzed (Participants) | 1 | 3 | 3 | 7
  %Transferrin Saturation Week 61: 50 - <69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 61: >=69: number analyzed (Participants) | 1 | 3 | 3 | 7
  %Transferrin Saturation Week 61: >=69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 73: <45: number analyzed (Participants) | 2 | 2 | 2 | 6
  %Transferrin Saturation Week 73: <45 | 2 | 1 | 2 | 5
  %Transferrin Saturation Week 73: 45 - <50: number analyzed (Participants) | 2 | 2 | 2 | 6
  %Transferrin Saturation Week 73: 45 - <50 | 0 | 1 | 0 | 1
  %Transferrin Saturation Week 73: 50 - <69: number analyzed (Participants) | 2 | 2 | 2 | 6
  %Transferrin Saturation Week 73: 50 - <69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 73: >=69: number analyzed (Participants) | 2 | 2 | 2 | 6
  %Transferrin Saturation Week 73: >=69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 85: <45: number analyzed (Participants) | 0 | 1 | 1 | 2
  %Transferrin Saturation Week 85: <45 | 0 | 1 | 1 | 2
  %Transferrin Saturation Week 85: 45 - <50: number analyzed (Participants) | 0 | 1 | 1 | 2
  %Transferrin Saturation Week 85: 45 - <50 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 85: 50 - <69: number analyzed (Participants) | 0 | 1 | 1 | 2
  %Transferrin Saturation Week 85: 50 - <69 | 0 | 0 | 0 | 0
  %Transferrin Saturation Week 85: >=69: number analyzed (Participants) | 0 | 1 | 1 | 2
  %Transferrin Saturation Week 85: >=69 | 0 | 0 | 0 | 0

14. Primary Outcome: Number of Participants With Significant Results of Physical Examinations Including Nose and Throat Mucosal Examinations
Description: Physical examinations were conducted by a physician, trained physician's assistant, or nurse practitioner as acceptable according to local regulation. A targeted nose and throat mucosal exam was performed to monitor for any signs of mucosal telangiectasias. The clinically significant physical examination results were determined by the investigator.
Time Frame: 2 Years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants | 0 | 0 | 0 | 0

15. Primary Outcome: Summary of Pubertal Development by Tanner Stage
Description: Tanner staging was performed before the first dose of this study to monitor for signs of accelerated sexual development. The physical changes in pubertal development (pubic hair, penis and testes) were assessed using the system described by Marshall and Tanner. Stage 1 is preadolescent, Stages 2, 3, and 4 are initiation of puberty and Stage 5 is mature adult. Details about the system can be referred to Tanner JM. Growth at Adolescence. Blackwell Scientific Publications 1962; 2nd edition.
  Participant's Week 97 visit within study B5161002 (parent study) was collected as screening data.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Screening, Baseline, Week 49.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Public Hair, Not Detected (ND) Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Public Hair, Not Detected (ND) Screening | 0 | 1 | 0 | 1
  Public Hair, Stage 1, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Public Hair, Stage 1, Screening | 1 | 0 | 0 | 1
  Public Hair, Stage 2, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Public Hair, Stage 2, Screening | 0 | 0 | 0 | 0
  Public Hair, Stage 3, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Public Hair, Stage 3, Screening | 0 | 0 | 0 | 0
  Public Hair, Stage 4, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Public Hair, Stage 4, Screening | 0 | 0 | 0 | 0
  Public Hair, Stage 5, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Public Hair, Stage 5, Screening | 0 | 0 | 0 | 0
  Public Hair, ND, Baseline | 1 | 0 | 0 | 1
  Public Hair, Stage 1, Baseline | 12 | 9 | 12 | 33
  Public Hair, Stage 2, Baseline | 5 | 10 | 8 | 23
  Public Hair, Stage 3, Baseline | 1 | 1 | 0 | 2
  Public Hair, Stage 4, Baseline | 0 | 0 | 0 | 0
  Public Hair, Stage 5, Baseline | 0 | 0 | 0 | 0
  Public Hair, ND/NA, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Public Hair, ND/NA, Week 49 | 0 | 0 | 0 | 0
  Public Hair, Stage 1, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Public Hair, Stage 1, Week 49 | 3 | 3 | 5 | 11
  Public Hair, Stage 2 Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Public Hair, Stage 2 Week 49 | 4 | 3 | 3 | 10
  Public Hair, Stage 3, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Public Hair, Stage 3, Week 49 | 0 | 0 | 0 | 0
  Public Hair, Stage 4, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Public Hair, Stage 4, Week 49 | 0 | 0 | 0 | 0
  Public Hair, Stage 5, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Public Hair, Stage 5, Week 49 | 0 | 0 | 0 | 0
  Penis, ND, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Penis, ND, Screening | 0 | 1 | 0 | 1
  Penis, Stage 1, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Penis, Stage 1, Screening | 1 | 0 | 0 | 1
  Penis, Stage 2, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Penis, Stage 2, Screening | 0 | 0 | 0 | 0
  Penis, Stage 3, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Penis, Stage 3, Screening | 0 | 0 | 0 | 0
  Penis, Stage 4, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Penis, Stage 4, Screening | 0 | 0 | 0 | 0
  Penis, Stage 5, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Penis, Stage 5, Screening | 0 | 0 | 0 | 0
  Penis, ND / NA, Baseline | 1 | 0 | 0 | 1
  Penis, Stage 1, Baseline | 13 | 11 | 11 | 35
  Penis, Stage 2, Baseline | 5 | 9 | 9 | 23
  Penis, Stage 3, Baseline | 0 | 0 | 0 | 0
  Penis, Stage 4, Baseline | 0 | 0 | 0 | 0
  Penis, Stage 5, Baseline | 0 | 0 | 0 | 0
  Penis, ND, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Penis, ND, Week 49 | 0 | 0 | 0 | 0
  Penis, Stage 1, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Penis, Stage 1, Week 49 | 4 | 2 | 4 | 10
  Penis, Stage 2, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Penis, Stage 2, Week 49 | 3 | 4 | 3 | 10
  Penis, Stage 3, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Penis, Stage 3, Week 49 | 0 | 0 | 1 | 1
  Penis, Stage 4, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Penis, Stage 4, Week 49 | 0 | 0 | 0 | 0
  Penis, Stage 5, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Penis, Stage 5, Week 49 | 0 | 0 | 0 | 0
  Testes, ND, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Testes, ND, Screening | 0 | 1 | 0 | 1
  Testes, Stage 1, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Testes, Stage 1, Screening | 1 | 0 | 0 | 1
  Testes, Stage 2, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Testes, Stage 2, Screening | 0 | 0 | 0 | 0
  Testes, Stage 3, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Testes, Stage 3, Screening | 0 | 0 | 0 | 0
  Testes, Stage 4, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Testes, Stage 4, Screening | 0 | 0 | 0 | 0
  Testes, Stage 5, Screening: number analyzed (Participants) | 1 | 1 | 0 | 2
  Testes, Stage 5, Screening | 0 | 0 | 0 | 0
  Testes, ND, Baseline | 1 | 0 | 0 | 1
  Testes, Stage 1, Baseline | 13 | 10 | 10 | 33
  Testes, Stage 2, Baseline | 5 | 9 | 10 | 24
  Testes, Stage 3, Baseline | 0 | 1 | 0 | 1
  Testes, Stage 4, Baseline | 0 | 0 | 0 | 0
  Testes, Stage 5, Baseline | 0 | 0 | 0 | 0
  Testes, ND, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Testes, ND, Week 49 | 0 | 0 | 0 | 0
  Testes, Stage 1, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Testes, Stage 1, Week 49 | 4 | 4 | 1 | 9
  Testes, Stage 2, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Testes, Stage 2, Week 49 | 3 | 2 | 6 | 11
  Testes, Stage 3, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Testes, Stage 3, Week 49 | 0 | 0 | 1 | 1
  Testes, Stage 4, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Testes, Stage 4, Week 49 | 0 | 0 | 0 | 0
  Testes, Stage 5, Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Testes, Stage 5, Week 49 | 0 | 0 | 0 | 0

16. Primary Outcome: Summary of Testicular Volume
Description: Testicular volume was used to monitor pubertal development. Participant's Week 97 visit within Study B5161002 (parent study) was collected as screening data in current study.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Screening, Baseline, Week 49.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 18 | 20 | 20 | 58
Milliliter
  Left Testis Volume - Screening: number analyzed (Participants) | 1 | 0 | 0 | 1
  Left Testis Volume - Screening | 3.0 (NA) — This was individual testicular volume. Standard deviation was not applicable. |  |  | 3.0 (NA) — This was individual testicular volume. Standard deviation was not applicable.
  Left Testis Volume - Baseline | 2.7 (1.07) | 2.8 (1.06) | 2.7 (1.63) | 2.7 (1.27)
  Left Testis Volume - Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Left Testis Volume - Week 49 | 2.6 (0.98) | 2.5 (0.55) | 3.8 (3.41) | 3.0 (2.19)
  Right Testis Volume - Screening: number analyzed (Participants) | 1 | 0 | 0 | 1
  Right Testis Volume - Screening | 3.0 (NA) — This was individual testicular volume. Standard deviation was not applicable. |  |  | 3.0 (NA) — This was individual testicular volume. Standard deviation was not applicable.
  Right Testis Volume - Baseline | 2.7 (1.03) | 2.8 (0.97) | 2.6 (1.64) | 2.7 (1.23)
  Right Testis Volume - Week 49: number analyzed (Participants) | 7 | 6 | 8 | 21
  Right Testis Volume - Week 49 | 2.6 (0.98) | 2.5 (0.55) | 3.6 (3.46) | 3.0 (2.20)

17. Primary Outcome: Number of Participants With Post-Baseline Vital Signs Data Meeting Categorical Summarization Criteria - B5161004 Baseline
Description: The number of participants pre-dose supine blood pressure and pulse rate meeting categorical summarization criteria are recorded in this table.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004.
  (DBP=diastolic blood pressure, SBP=systolic blood pressure; The unit for blood pressure is: mmHg, the unit for pulse rate is: beats per minute [BPM])
Time Frame: 2 Years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Supine SBP - Observed Values <70+2×Age (2-10years): number analyzed (Participants) | 17 | 12 | 6 | 35
  Supine SBP - Observed Values <70+2×Age (2-10years) | 1 | 1 | 0 | 2
  Supine SBP - Observed Values < 90 (11-17 years): number analyzed (Participants) | 2 | 8 | 14 | 24
  Supine SBP - Observed Values < 90 (11-17 years) | 0 | 1 | 1 | 2
  Maximum Increase From Baseline in Supine SBP >=30 | 1 | 0 | 3 | 4
  Maximum Decrease From Baseline in Supine SBP >=30 | 0 | 1 | 0 | 1
  Supine DBP - Observed Values <50 (<18 years) | 1 | 1 | 2 | 4
  Maximum Increase From Baseline in Supine DBP >=20 | 3 | 1 | 5 | 9
  Maximum Decrease From Baseline in Supine DBP >=20 | 0 | 2 | 0 | 2
  Supine Pulse Rate-Observed Values<40BPM(<18 years) | 0 | 0 | 0 | 0
  Supine Pulse Rate-Observed Values>120BPM(<18years) | 2 | 0 | 1 | 3

18. Primary Outcome: Number of Participants With Post-Baseline Vital Signs Data Meeting Categorical Summarization Criteria - Overall Baseline
Description: The number of participants with data of pre-dose supine blood pressure meeting categorical summarization were recorded in this table.
  Overall Baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002.
  (DBP=diastolic blood pressure, SBP=systolic blood pressure; The unit for blood pressure is: mmHg).
Time Frame: 2 Years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Maximum Increase From Baseline in Supine SBP >=30 | 2 | 6 | 2 | 10
  Maximum Decrease From Baseline in Supine SBP >=30 | 0 | 3 | 4 | 7
  Maximum Increase From Baseline in Supine DBP >=20 | 8 | 8 | 10 | 26
  Maximum Decrease From Baseline in Supine DBP >=20 | 4 | 4 | 8 | 16

19. Primary Outcome: Number of Participants With Post-Baseline ECG Data Meeting Categorical Summarization Criteria - B5161004 Baseline
Description: QTcF=QT/(60/Hour)**(1/3). Means of replicates were used in the calculations. QT=time between the start of the Q wave and the end of the T wave in the heart's electrical cycle; QTcF=corrected QT (Fridericia correction). All scheduled ECGs were performed after the participant had rested quietly for at least 10 minutes in a supine position.
  Baseline was defined as the average of the last triplicate pre-dose measurements prior to Day 1 in B5161004.
Time Frame: 2 Years
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 18 | 20 | 20 | 58
Participants
  Maximum(Max)QTcF Interval-ObservedValues<450msec | 18 | 20 | 18 | 56
  Max QTcF Interval -Observed Values450-<480msec | 0 | 0 | 2 | 2
  Max QTcF Interval -Observed Values480-<500msec | 0 | 0 | 0 | 0
  Max QTcF Interval -Observed Values>=500msec | 0 | 0 | 0 | 0
  Max QTcF Interval Increase From Baseline<30msec | 16 | 20 | 18 | 54
  Max QTcF Interval Increase From Baseline30-<60msec | 2 | 0 | 0 | 2
  Max QTcF Interval Increase From Baseline>= 60msec | 0 | 0 | 2 | 2

20. Primary Outcome: Number of Participants With Post-Baseline ECG Data Meeting Categorical Summarization Criteria - Overall Baseline
Description: QT=time between the start of the Q wave and the end of the T wave in the heart's electrical cycle; QTcF=corrected QT (Fridericia correction). All scheduled ECGs were performed after the participant had rested quietly for at least 10 minutes in a supine position.
  Overall baseline was defined as the average of the last triplicate pre-dose measurements prior to the first day of dosing in study B5161002.
Time Frame: 2 Years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Maximum QTcF Interval Increase From Baseline <30 | 11 | 15 | 17 | 43
  Max-QTcF Interval IncreaseFromBaseline30-<60msec | 7 | 5 | 1 | 13
  Maximum QTcF Interval Increase From Baseline >=60 | 1 | 0 | 2 | 3

21. Primary Outcome: Number of Participants With Iron Accumulation Data Meeting Categorical Summarization Criteria
Description: Liver Magnetic Resonance Imaging (MRIs) were sent to an independent central radiology imaging facility for calculation of the average R2* value which was used to monitor for iron accumulation in the liver. Mean R2* values had been used in the calculations.
  Normal: R2* <= 75 Hz at 1.5 T or <=139 Hz at 3.0 T; Above Normal: R2* > 75 Hz and <= 190 Hz at 1.5 T or R2* > 139 Hz and <= 369 Hz at 3.0 T Mild overload: R2* > 190 Hz at 1.5 T or R2* > 369 Hz at 3.0 T Data from participant's Week 93 visit in Study B5161002 (parent study) were used for screening in the current study.
Time Frame: Screening and Week 49.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Screening - Normal | 19 | 20 | 20 | 59
  Screening - Above Normal | 0 | 0 | 0 | 0
  Screening - Mild Overload | 0 | 0 | 0 | 0
  Week 49 - Normal: number analyzed (Participants) | 7 | 6 | 8 | 21
  Week 49 - Normal | 7 | 6 | 8 | 21
  Week 49 - Above Normal: number analyzed (Participants) | 7 | 6 | 8 | 21
  Week 49 - Above Normal | 0 | 0 | 0 | 0
  Week 49 - Mild Overload: number analyzed (Participants) | 7 | 6 | 8 | 21
  Week 49 - Mild Overload | 0 | 0 | 0 | 0
  Total - Normal | 19 | 20 | 20 | 59
  Total - Above Normal | 0 | 0 | 0 | 0
  Total - Mild Overload | 0 | 0 | 0 | 0

22. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) by Cardiac MRI - B5161004 Baseline
Description: The LVEF was the ratio of blood ejected during systole to blood in the ventricle at the end of diastole. LVEF was measured by cardiac magnetic resonance imaging (MRI) or echocardiography. The same method of cardiac imaging was used consistently for each participant. Cardiac MRIs were read by a central imaging vendor, while echocardiograms were read locally (at each site). The table presents the results from cardiac MRIs. Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline and Week 49.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio of Ejected Blood
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Ratio of Ejected Blood
  Baseline - Observed Values: number analyzed (Participants) | 2 | 4 | 5 | 11
  Baseline - Observed Values | 56.000 (5.6569) | 60.750 (2.2174) | 62.400 (5.6833) | 60.636 (4.8430)
  Week 49 - Change From Baseline: number analyzed (Participants) | 1 | 0 | 2 | 3
  Week 49 - Change From Baseline | -3.000 (NA) — Standard deviation was not applicable for individual value. |  | -1.500 (4.9497) | -2.000 (3.6056)

23. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) by Cardiac MRI - Overall Baseline
Description: The LVEF was the ratio of blood ejected during systole to blood in the ventricle at the end of diastole. LVEF was measured by cardiac magnetic resonance imaging (MRI) or echocardiography. The same method of cardiac imaging was used consistently for each participant. Cardiac MRIs were read by a central imaging vendor, while echocardiograms were read locally (at each site). The table presents the results from cardiac MRIs.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was counted starting from the study treatment in study B5161002.
Time Frame: Baseline, Weeks 49, 97, 146.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio of Ejected Blood
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Ratio of Ejected Blood
  Baseline - Observed Values: number analyzed (Participants) | 2 | 4 | 6 | 12
  Baseline - Observed Values | 66.000 (8.4853) | 61.250 (3.5000) | 61.333 (5.3541) | 62.083 (5.1250)
  Week 49 - Change From Baseline: number analyzed (Participants) | 2 | 4 | 5 | 11
  Week 49 - Change From Baseline | -11.000 (2.8284) | -3.500 (1.9149) | 0.000 (7.4498) | -3.273 (6.4357)
  Week 97 - Change From Baseline: number analyzed (Participants) | 2 | 4 | 5 | 11
  Week 97 - Change From Baseline | -10.000 (2.8284) | -0.500 (2.8868) | -0.800 (6.5727) | -2.364 (5.9038)
  Week 146 - Change From Baseline: number analyzed (Participants) | 1 | 0 | 2 | 3
  Week 146 - Change From Baseline | -15.000 (NA) — Standard deviation was not applicable for individual value. |  | 3.500 (0.7071) | -2.667 (10.6927)

24. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) by Echocardiogram - B5161004 Baseline
Description: The LVEF was the ratio of blood ejected during systole to blood in the ventricle at the end of diastole. LVEF was measured by cardiac magnetic resonance imaging (MRI) or echocardiography. The same method of cardiac imaging was used consistently for each participant. Cardiac MRIs were read by a central imaging vendor, while echocardiograms were read locally (at each site). The table presents the results from echocardiograms.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Week 49.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio of Ejected Blood
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Ratio of Ejected Blood
  Baseline - Observed Values: number analyzed (Participants) | 17 | 17 | 14 | 48
  Baseline - Observed Values | 60.359 (3.7545) | 62.461 (6.0180) | 62.543 (5.3731) | 61.740 (5.1170)
  Week 49 - Change From Baseline: number analyzed (Participants) | 5 | 6 | 5 | 16
  Week 49 - Change From Baseline | -0.400 (5.0334) | -3.900 (8.9252) | 2.200 (7.6056) | -0.900 (7.4580)

25. Primary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) by Echocardiogram - Overall Baseline
Description: The LVEF was the ratio of blood ejected during systole to blood in the ventricle at the end of diastole. LVEF was measured by cardiac magnetic resonance imaging (MRI) or echocardiography. The same method of cardiac imaging was used consistently for each participant. Cardiac MRIs were read by a central imaging vendor, while echocardiograms were read locally (at each site). The table presents the results from echocardiograms.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was counted starting from the study treatment in study B5161002.
Time Frame: Baseline, Weeks 49, 97, 146.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio of Ejected Blood
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Ratio of Ejected Blood
  Baseline - Observed Values: number analyzed (Participants) | 17 | 16 | 15 | 48
  Baseline - Observed Values | 63.288 (4.3743) | 64.094 (4.3025) | 64.073 (4.5848) | 63.802 (4.3395)
  Week 49 - Change From Baseline: number analyzed (Participants) | 17 | 15 | 15 | 47
  Week 49 - Change From Baseline | -0.171 (5.7432) | -1.040 (4.8861) | -0.213 (6.1487) | -0.462 (5.5142)
  Week 97 - Change From Baseline: number analyzed (Participants) | 17 | 16 | 14 | 47
  Week 97 - Change From Baseline | -2.929 (5.4060) | -1.810 (6.1321) | -1.414 (6.4799) | -2.097 (5.8924)
  Week 146 - Change From Baseline: number analyzed (Participants) | 5 | 6 | 5 | 16
  Week 146 - Change From Baseline | -1.240 (2.3416) | -4.833 (4.2151) | -1.440 (11.6993) | -2.650 (6.8514)

26. Primary Outcome: Bone Age to Chronological Age Ratio
Description: Bone age assessment was evaluated by the ratio of the bone age to the chronological age using the X rays of the hand and wrist. Ratio of bone age to chronological age was calculated by bone age/chronological age at scan date. Chronological age at scan date was calculated by (scan date - date of birth + 1)/365.25.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline and Week 49.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Ratio
  Baseline | 0.76 (0.213) | 0.74 (0.195) | 0.81 (0.177) | 0.77 (0.194)
  Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Week 49 | 0.74 (0.197) | 0.65 (0.157) | 0.70 (0.172) | 0.70 (0.172)

27. Primary Outcome: Whole Body and Spine DXA: Bone Mineral Density Z-Score, Height Adjusted Over Time
Description: Bone mineral density (BMD) was monitored by dual energy x-ray absorptiometry (DXA). DXA scans were obtained to evaluate bone mineral density of the spine and whole body without head.
  The height adjusted Z-score presented below is the number of standard deviations which compares the BMD of the participant to the average BMD matched for their age, sex and ethnicity. If the Z-score was -2 standard deviations or lower, the result was "below the expected range for age". If the Z-score was above -2 standard deviations, the result was "within the expected range for age".
Time Frame: Screening (Week 97 visit within parent study B5161002) and Week 49
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Standard Deviations
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Standard Deviations
  Anterior Posterior Spine Total L1 to L4 -Screening: number analyzed (Participants) | 18 | 20 | 16 | 54
  Anterior Posterior Spine Total L1 to L4 -Screening | -0.687659 (0.9152662) | -0.587384 (1.0241266) | -0.561789 (1.0285799) | -0.613225 (0.9731687)
  Anterior Posterior Spine Total L1 to L4 - Week 49: number analyzed (Participants) | 7 | 5 | 5 | 17
  Anterior Posterior Spine Total L1 to L4 - Week 49 | -0.131374 (0.9251749) | -0.435384 (0.5747293) | -0.152854 (1.7877768) | -0.227106 (1.1053887)
  Body Without Head - Screening | -1.936367 (1.1544544) | -1.956332 (1.3561294) | -1.872619 (1.4843432) | -1.921525 (1.3187696)
  Body Without Head - Week 49: number analyzed (Participants) | 7 | 6 | 6 | 19
  Body Without Head - Week 49 | -1.789347 (1.1738270) | -1.943538 (1.6839551) | -1.455670 (1.5655008) | -1.732667 (1.4033563)

28. Primary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) was performed to identify the risk of suicide ideation or behavior. C-SSRS was conducted with the participant's caregiver/legal guardian on the participant's behalf throughout the study, rather than administering this evaluation directly with the study participants. If at any visit the participant endorsed a 4 or 5 on the C-SSRS ideation section or reported any suicidality behavior, then an evaluation of suicide risk (risk assessment) had to be completed and the participant must have been discontinued. The significant result of C-SSRS was determined by the investigator.
Time Frame: 2 Years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Suicidal Ideation | 0 | 0 | 0 | 0
  Suicidal Behavior | 0 | 0 | 0 | 0

29. Secondary Outcome: Change From Baseline on the 4 Stair Climb (4SC) - B5161004 Baseline
Description: The 4SC quantified the time required for a participant to ascend 4 standard steps. The functional assessment of 4SC was conducted by a physiotherapist (or exercise physiologist). In order to provide optimal testing conditions and consistency in endpoint measurements, the functional assessments were completed at approximately the same time of day.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49, 73.
Population: This analysis population included all participants who had received at least 1 dose of study medication in current study B5161004.
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Seconds
  Baseline: number analyzed (Participants) | 15 | 13 | 11 | 39
  Baseline | 7.268 [3.779 to 10.757] | 5.218 [3.370 to 7.065] | 5.373 [2.936 to 7.809] | 6.050 [4.530 to 7.570]
  Week 13: number analyzed (Participants) | 15 | 13 | 11 | 39
  Week 13 | 0.839 [-0.680 to 2.357] | 0.821 [0.178 to 1.463] | 0.400 [-0.416 to 1.216] | 0.709 [0.098 to 1.320]
  Week 25: number analyzed (Participants) | 10 | 9 | 8 | 27
  Week 25 | 1.248 [-0.050 to 2.546] | 0.319 [-0.073 to 0.710] | 0.663 [-0.368 to 1.693] | 0.765 [0.236 to 1.294]
  Week 49: number analyzed (Participants) | 6 | 4 | 5 | 15
  Week 49 | 10.150 [-5.363 to 25.663] | 0.998 [-0.140 to 2.135] | 2.400 [-2.917 to 7.717] | 5.126 [-0.460 to 10.712]
  Week 73: number analyzed (Participants) | 2 | 2 | 1 | 5
  Week 73 | 9.350 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 3.100 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 1.000 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 5.180 [-0.234 to 10.594]

30. Secondary Outcome: Change From Baseline on the 4SC - Overall Baseline
Description: The 4SC quantified the time required for a participant to ascend 4 standard steps. The functional assessment of 4SC was conducted by a physiotherapist (or exercise physiologist). In order to provide optimal testing conditions and consistency in endpoint measurements, the functional assessments were completed at approximately the same time of day.
  This is the overall change from baseline which included the change since enrolling in the parent study B5161002.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was counted starting from the study treatment in study B5161002.
Time Frame: Baseline, Weeks 9,17,25,33,41,49,57,65,73,81,89,97,110,122,146,170.
Population: The analysis population included all participants who had received at least 1 dose of study medication in current study B5161004. Number of participants analyzed signifies number of participants who were evaluable for this outcome measure. Number analyzed refers to number of participants evaluable for specified rows of categories.
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Seconds
  Baseline | 4.381 [3.442 to 5.319] | 5.664 [3.728 to 7.599] | 5.717 [4.141 to 7.292] | 5.268 [4.409 to 6.128]
  Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Week 9 | -0.096 [-0.582 to 0.389] | 0.898 [-0.444 to 2.240] | 0.879 [0.103 to 1.654] | 0.566 [0.046 to 1.085]
  Week 17: number analyzed (Participants) | 19 | 17 | 19 | 55
  Week 17 | 0.500 [-0.365 to 1.365] | 2.270 [-0.898 to 5.438] | 1.493 [0.009 to 2.977] | 1.390 [0.309 to 2.472]
  Week 25: number analyzed (Participants) | 18 | 18 | 17 | 53
  Week 25 | 0.427 [-0.385 to 1.239] | 2.835 [0.094 to 5.576] | 2.836 [-0.775 to 6.447] | 2.018 [0.577 to 3.458]
  Week 33: number analyzed (Participants) | 18 | 18 | 17 | 53
  Week 33 | 1.298 [-1.043 to 3.639] | 3.713 [-0.573 to 7.999] | 1.804 [0.151 to 3.457] | 2.280 [0.630 to 3.930]
  Week 41: number analyzed (Participants) | 18 | 17 | 16 | 51
  Week 41 | 0.920 [-0.665 to 2.505] | 3.361 [-1.170 to 7.892] | 2.217 [0.192 to 4.241] | 2.140 [0.508 to 3.773]
  Week 49: number analyzed (Participants) | 17 | 16 | 16 | 49
  Week 49 | 0.480 [-0.040 to 1.000] | 2.391 [0.151 to 4.630] | 1.898 [0.397 to 3.399] | 1.567 [0.704 to 2.430]
  Week 57: number analyzed (Participants) | 17 | 16 | 14 | 47
  Week 57 | 0.712 [0.129 to 1.294] | 3.827 [-0.137 to 7.791] | 2.914 [-0.289 to 6.118] | 2.428 [0.846 to 4.010]
  Week 65: number analyzed (Participants) | 17 | 16 | 12 | 45
  Week 65 | 1.337 [0.141 to 2.533] | 4.259 [0.138 to 8.380] | 2.181 [-1.064 to 5.426] | 2.601 [0.941 to 4.261]
  Week 73: number analyzed (Participants) | 16 | 15 | 14 | 45
  Week 73 | 1.561 [0.066 to 3.055] | 3.082 [0.752 to 5.412] | 1.849 [0.178 to 3.520] | 2.157 [1.150 to 3.164]
  Week 81: number analyzed (Participants) | 16 | 14 | 14 | 44
  Week 81 | 1.633 [0.561 to 2.704] | 3.006 [-0.084 to 6.096] | 2.262 [-0.026 to 4.550] | 2.270 [1.087 to 3.453]
  Week 89: number analyzed (Participants) | 17 | 13 | 13 | 43
  Week 89 | 1.687 [0.680 to 2.694] | 2.069 [0.779 to 3.359] | 3.182 [-0.296 to 6.661] | 2.255 [1.161 to 3.349]
  Week 97: number analyzed (Participants) | 17 | 13 | 13 | 43
  Week 97 | 2.652 [0.323 to 4.981] | 1.874 [0.562 to 3.185] | 1.790 [0.217 to 3.363] | 2.156 [1.123 to 3.189]
  Week 110: number analyzed (Participants) | 15 | 13 | 11 | 39
  Week 110 | 3.811 [0.071 to 7.552] | 2.748 [0.950 to 4.547] | 1.806 [-0.435 to 4.048] | 2.892 [1.330 to 4.453]
  Week 122: number analyzed (Participants) | 10 | 9 | 8 | 27
  Week 122 | 3.128 [0.653 to 5.603] | 1.781 [0.760 to 2.802] | 1.909 [-0.412 to 4.229] | 2.318 [1.259 to 3.377]
  Week 146: number analyzed (Participants) | 6 | 4 | 5 | 15
  Week 146 | 11.933 [-4.591 to 28.458] | 2.498 [-1.975 to 6.970] | 4.034 [-3.016 to 11.084] | 6.784 [0.749 to 12.819]
  Week 170: number analyzed (Participants) | 2 | 2 | 1 | 5
  Week 170 | 10.450 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 6.150 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 2.100 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 7.060 [1.542 to 12.578]

31. Secondary Outcome: Change From Baseline on the Forced Vital Capacity (FVC) - B5161004 Baseline
Description: FVC was measured using the FVC maneuver by spirometry to evaluate respiratory muscle function. The best (largest) FVC measurement from a set of 3 was captured on the database.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49 and 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Litres
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Litres
  Baseline: number analyzed (Participants) | 16 | 17 | 18 | 51
  Baseline | 1.6550 [1.4829 to 1.8271] | 1.7029 [1.4607 to 1.9452] | 1.8678 [1.6245 to 2.1110] | 1.7461 [1.6227 to 1.8694]
  Week 13: number analyzed (Participants) | 16 | 16 | 15 | 47
  Week 13 | 0.0344 [-0.0355 to 0.1042] | 0.1106 [-0.0620 to 0.2832] | 0.0380 [-0.0417 to 0.1177] | 0.0615 [-0.0024 to 0.1254]
  Week 25: number analyzed (Participants) | 11 | 12 | 14 | 37
  Week 25 | 0.0718 [-0.0701 to 0.2137] | 0.1467 [0.0081 to 0.2852] | 0.1086 [-0.0094 to 0.2266] | 0.1100 [0.0409 to 0.1791]
  Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Week 49 | 0.2086 [0.0862 to 0.3310] | 0.2633 [-0.0621 to 0.5887] | 0.0671 [-0.0385 to 0.1728] | 0.1755 [0.0794 to 0.2716]
  Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Week 73 | 0.2800 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.3750 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.1450 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.2667 [-0.0373 to 0.5707]

32. Secondary Outcome: Change From Baseline on the FVC - Overall Baseline
Description: Forced vital capacity (FVC) was measured using the FVC maneuver by spirometry to evaluate respiratory muscle function. The best (largest) FVC measurement from a set of 3 was captured on the database. This is the overall change from baseline which included the change since enrolling in the parent study B5161002.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was counted starting from the study treatment in study B5161002.
Time Frame: Baseline, Weeks 9,17,25,33,41,49,57,65,73,81,89,97,110,122,146,170.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Litres
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Litres
  Baseline | 1.3753 [1.2305 to 1.5200] | 1.5810 [1.4256 to 1.7364] | 1.6265 [1.4322 to 1.8208] | 1.5302 [1.4353 to 1.6250]
  Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Week 9 | 0.1205 [0.0093 to 0.2317] | 0.1089 [-0.0307 to 0.2486] | -0.0435 [-0.1331 to 0.0461] | 0.0602 [-0.0049 to 0.1253]
  Week 17 | 0.0837 [-0.0234 to 0.1907] | 0.0700 [-0.0113 to 0.1513] | 0.0585 [-0.0097 to 0.1267] | 0.0705 [0.0237 to 0.1173]
  Week 25 | 0.0679 [-0.0461 to 0.1819] | 0.1140 [0.0204 to 0.2076] | -0.0135 [-0.1276 to 0.1006] | 0.0559 [-0.0040 to 0.1158]
  Week 33 | 0.1463 [0.0379 to 0.2548] | 0.0740 [-0.0414 to 0.1894] | 0.1100 [0.0425 to 0.1775] | 0.1095 [0.0553 to 0.1637]
  Week 41 | 0.1484 [0.0343 to 0.2625] | 0.1115 [-0.0298 to 0.2528] | 0.1320 [0.0582 to 0.2058] | 0.1303 [0.0689 to 0.1918]
  Week 49: number analyzed (Participants) | 18 | 20 | 20 | 58
  Week 49 | 0.1328 [-0.0053 to 0.2709] | 0.1350 [0.0427 to 0.2273] | 0.1565 [0.1011 to 0.2119] | 0.1417 [0.0886 to 0.1948]
  Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Week 57 | 0.1063 [-0.0470 to 0.2597] | 0.1735 [0.0607 to 0.2863] | 0.1656 [0.0406 to 0.2905] | 0.1486 [0.0772 to 0.2200]
  Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Week 65 | 0.2005 [0.0530 to 0.3480] | 0.1830 [0.0959 to 0.2701] | 0.1726 [0.0647 to 0.2806] | 0.1853 [0.1225 to 0.2482]
  Week 73: number analyzed (Participants) | 18 | 20 | 20 | 58
  Week 73 | 0.1706 [-0.0177 to 0.3588] | 0.1925 [0.0706 to 0.3144] | 0.1330 [0.0521 to 0.2139] | 0.1652 [0.0927 to 0.2376]
  Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Week 81 | 0.2263 [0.0718 to 0.3808] | 0.1353 [0.0110 to 0.2595] | 0.2045 [0.1279 to 0.2811] | 0.1890 [0.1225 to 0.2554]
  Week 89: number analyzed (Participants) | 17 | 20 | 20 | 57
  Week 89 | 0.2406 [0.0674 to 0.4137] | 0.1960 [0.0389 to 0.3531] | 0.2145 [0.1087 to 0.3203] | 0.2158 [0.1369 to 0.2946]
  Week 97 | 0.2932 [0.1616 to 0.4247] | 0.1365 [-0.0336 to 0.3066] | 0.2375 [0.1472 to 0.3278] | 0.2212 [0.1462 to 0.2962]
  Week 110: number analyzed (Participants) | 16 | 16 | 15 | 47
  Week 110 | 0.2781 [0.1373 to 0.4189] | 0.2256 [0.0736 to 0.3777] | 0.2407 [0.1167 to 0.3646] | 0.2483 [0.1734 to 0.3232]
  Week 122: number analyzed (Participants) | 11 | 12 | 14 | 37
  Week 122 | 0.2973 [0.0532 to 0.5413] | 0.3708 [0.2666 to 0.4750] | 0.3221 [0.1436 to 0.5007] | 0.3305 [0.2360 to 0.4250]
  Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Week 146 | 0.4629 [0.1599 to 0.7658] | 0.4167 [0.1726 to 0.6607] | 0.3114 [0.1531 to 0.4698] | 0.3960 [0.2797 to 0.5123]
  Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Week 170 | 0.5500 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.2850 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.4900 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.4417 [0.1950 to 0.6884]

33. Secondary Outcome: Change From Baseline on the Northstar Ambulatory Assessment (NSAA) Score - B5161004 Baseline
Description: The NSAA was a 17-item test that measured gross motor function. Each individual item was evaluated with either 0-unable to perform independently, 1-able to perform with assistance, 2-able to perform without assistance. A total score was achieved by summing all the individual items. The total score could range from 0 to 34 (fully-independent function).
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49, 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Units on a Scale
  Baseline: number analyzed (Participants) | 15 | 17 | 17 | 49
  Baseline | 16.4 [11.8 to 21.0] | 17.1 [11.6 to 22.6] | 12.9 [6.9 to 19.0] | 15.4 [12.5 to 18.4]
  Week 13: number analyzed (Participants) | 15 | 17 | 16 | 48
  Week 13 | -0.6 [-1.3 to 0.1] | -1.7 [-3.0 to -0.4] | -0.4 [-1.6 to 0.7] | -0.9 [-1.5 to -0.3]
  Week 25: number analyzed (Participants) | 10 | 12 | 13 | 35
  Week 25 | -1.8 [-3.1 to -0.5] | -0.7 [-1.6 to 0.2] | -0.8 [-2.0 to 0.5] | -1.0 [-1.7 to -0.4]
  Week 49: number analyzed (Participants) | 7 | 6 | 6 | 19
  Week 49 | -3.6 [-6.9 to -0.2] | -3.2 [-5.8 to -0.6] | -3.2 [-5.6 to -0.7] | -3.3 [-4.6 to -2.0]
  Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Week 73 | -5.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -3.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -4.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -4.2 [-7.4 to -1.0]

34. Secondary Outcome: Change From Baseline on the NSAA Score - Overall Baseline
Description: The NSAA was a 17-item test that measured gross motor function. Each individual item was evaluated with either 0-unable to perform independently, 1-able to perform with assistance, 2-able to perform without assistance. A total score was achieved by summing all the individual items. The total score could range from 0 to 34 (fully-independent function). This is the overall change from baseline which included the change since enrolling in the parent study B5161002.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was counted starting from the study treatment in study B5161002.
Time Frame: Baseline, Weeks 9,17,25,33,41,49,57,65,73,81,89,97,110,122,146,170.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Units on a Scale
  Baseline | 20.8 [17.6 to 24.1] | 21.2 [17.2 to 25.2] | 19.5 [16.0 to 23.0] | 20.5 [18.5 to 22.5]
  Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Week 9 | -0.2 [-1.3 to 1.0] | 0.4 [-0.6 to 1.4] | -0.8 [-2.4 to 0.8] | -0.2 [-0.9 to 0.5]
  Week 17: number analyzed (Participants) | 19 | 20 | 19 | 58
  Week 17 | 0.3 [-1.1 to 1.6] | -2.2 [-5.8 to 1.5] | -0.9 [-2.7 to 0.9] | -0.9 [-2.3 to 0.4]
  Week 25 | 0.1 [-1.5 to 1.7] | -1.4 [-3.1 to 0.3] | -2.2 [-4.7 to 0.4] | -1.2 [-2.3 to 0.0]
  Week 33 | -0.4 [-2.0 to 1.2] | -1.5 [-3.1 to 0.1] | -2.9 [-5.1 to -0.7] | -1.6 [-2.7 to -0.6]
  Week 41 | -1.5 [-3.8 to 0.7] | -2.7 [-4.5 to -0.8] | -3.6 [-6.0 to -1.2] | -2.6 [-3.8 to -1.4]
  Week 49: number analyzed (Participants) | 19 | 20 | 19 | 58
  Week 49 | -1.8 [-4.2 to 0.6] | -3.4 [-5.5 to -1.2] | -4.2 [-6.9 to -1.6] | -3.1 [-4.5 to -1.8]
  Week 57: number analyzed (Participants) | 18 | 20 | 19 | 57
  Week 57 | -2.6 [-5.1 to -0.2] | -3.7 [-6.0 to -1.3] | -5.5 [-9.3 to -1.6] | -3.9 [-5.6 to -2.3]
  Week 65: number analyzed (Participants) | 18 | 20 | 20 | 58
  Week 65 | -2.7 [-5.4 to -0.1] | -3.8 [-6.1 to -1.5] | -5.8 [-9.6 to -1.9] | -4.1 [-5.8 to -2.5]
  Week 73: number analyzed (Participants) | 18 | 20 | 20 | 58
  Week 73 | -4.7 [-7.7 to -1.6] | -5.1 [-7.4 to -2.7] | -5.8 [-8.8 to -2.7] | -5.2 [-6.7 to -3.6]
  Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Week 81 | -4.1 [-6.8 to -1.3] | -4.5 [-6.9 to -2.1] | -6.0 [-9.3 to -2.6] | -4.9 [-6.4 to -3.3]
  Week 89: number analyzed (Participants) | 18 | 19 | 20 | 57
  Week 89 | -4.2 [-7.5 to -1.0] | -6.2 [-8.5 to -3.9] | -7.4 [-10.4 to -4.3] | -6.0 [-7.6 to -4.4]
  Week 97: number analyzed (Participants) | 18 | 20 | 20 | 58
  Week 97 | -4.4 [-7.7 to -1.1] | -6.7 [-9.3 to -4.0] | -7.0 [-10.0 to -3.9] | -6.1 [-7.7 to -4.4]
  Week 110: number analyzed (Participants) | 16 | 17 | 16 | 49
  Week 110 | -5.1 [-8.4 to -1.8] | -7.2 [-9.8 to -4.7] | -5.9 [-8.9 to -2.9] | -6.1 [-7.7 to -4.5]
  Week 122: number analyzed (Participants) | 11 | 12 | 13 | 36
  Week 122 | -6.4 [-11.7 to -1.0] | -7.2 [-10.7 to -3.6] | -7.6 [-12.0 to -3.3] | -7.1 [-9.4 to -4.8]
  Week 146: number analyzed (Participants) | 7 | 6 | 6 | 19
  Week 146 | -9.9 [-19.7 to 0.0] | -8.3 [-13.2 to -3.5] | -7.3 [-10.1 to -4.5] | -8.6 [-11.9 to -5.3]
  Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Week 170 | -11.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -12.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -7.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -10.2 [-15.6 to -4.8]

35. Secondary Outcome: Change From Baseline on the NSAA - Time to Stand From Supine - B5161004 Baseline
Description: Rise from supine was a timed functional test within NSAA. This test of time-to-stand from supine was analyzed separately for summary tabulation along with the total NSAA score.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49, 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Seconds
  Baseline: number analyzed (Participants) | 6 | 11 | 8 | 25
  Baseline | 4.517 [2.612 to 6.421] | 6.508 [3.996 to 9.020] | 6.250 [4.552 to 7.948] | 5.948 [4.751 to 7.144]
  Week 13: number analyzed (Participants) | 6 | 11 | 8 | 25
  Week 13 | 0.330 [-0.231 to 0.891] | 1.353 [0.357 to 2.349] | -0.038 [-0.931 to 0.856] | 0.662 [0.121 to 1.203]
  Week 25: number analyzed (Participants) | 4 | 8 | 6 | 18
  Week 25 | -0.113 [-0.585 to 0.360] | 1.463 [0.315 to 2.610] | -0.167 [-1.410 to 1.076] | 0.569 [-0.112 to 1.251]
  Week 49: number analyzed (Participants) | 1 | 4 | 4 | 9
  Week 49 | 0.670 [NA to NA] — 95% Confidence Interval was not applicable for individual value. | 1.518 [-1.384 to 4.419] | 2.978 [-1.944 to 7.899] | 2.072 [0.246 to 3.898]
  Week 73: number analyzed (Participants) | 0 | 1 | 1 | 2
  Week 73 |  | 10.170 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 2.300 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 6.235 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval.

36. Secondary Outcome: Change From Baseline on the NSAA - Time to Stand From Supine - Overall Baseline
Description: Rise from supine was a timed functional test within NSAA. This test of time-to-stand from supine was analyzed separately for summary tabulation along with the total NSAA score. This is the overall change from baseline which included the change since enrolling in the parent study B5161002.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was counted starting from the study treatment in study B5161002.
Time Frame: Baseline, Weeks 9,17,25,33,41,49,57,65,73,81,89,97,110,122,146,170.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Seconds
  Baseline: number analyzed (Participants) | 16 | 15 | 15 | 46
  Baseline | 6.440 [4.446 to 8.434] | 7.059 [2.997 to 11.122] | 7.046 [5.130 to 8.962] | 6.840 [5.348 to 8.331]
  Week 9: number analyzed (Participants) | 16 | 14 | 12 | 42
  Week 9 | -0.140 [-1.049 to 0.769] | 0.486 [-0.190 to 1.163] | 0.867 [-0.101 to 1.834] | 0.356 [-0.116 to 0.829]
  Week 17: number analyzed (Participants) | 16 | 12 | 13 | 41
  Week 17 | 10.251 [-11.639 to 32.142] | 1.123 [0.185 to 2.060] | 1.148 [0.013 to 2.282] | 4.693 [-3.384 to 12.770]
  Week 25: number analyzed (Participants) | 16 | 12 | 10 | 38
  Week 25 | 1.283 [-0.135 to 2.701] | 0.514 [0.055 to 0.973] | 1.456 [-0.401 to 3.313] | 1.086 [0.364 to 1.808]
  Week 33: number analyzed (Participants) | 15 | 12 | 11 | 38
  Week 33 | 1.382 [-0.038 to 2.802] | 0.392 [-0.412 to 1.195] | 1.143 [-1.200 to 3.485] | 1.000 [0.166 to 1.834]
  Week 41: number analyzed (Participants) | 14 | 12 | 10 | 36
  Week 41 | 1.184 [0.123 to 2.246] | 0.526 [-0.230 to 1.282] | 1.620 [-0.213 to 3.453] | 1.086 [0.445 to 1.726]
  Week 49: number analyzed (Participants) | 14 | 12 | 12 | 38
  Week 49 | 1.642 [-0.005 to 3.289] | 0.730 [-0.466 to 1.926] | 1.630 [0.269 to 2.991] | 1.350 [0.582 to 2.118]
  Week 57: number analyzed (Participants) | 13 | 11 | 9 | 33
  Week 57 | 1.577 [-0.212 to 3.366] | 1.376 [-0.184 to 2.937] | 1.316 [-0.581 to 3.212] | 1.439 [0.534 to 2.343]
  Week 65: number analyzed (Participants) | 12 | 11 | 9 | 32
  Week 65 | 1.590 [-0.715 to 3.895] | 1.570 [-0.113 to 3.253] | 1.907 [-0.652 to 4.465] | 1.672 [0.556 to 2.788]
  Week 73: number analyzed (Participants) | 12 | 11 | 11 | 34
  Week 73 | 2.664 [0.149 to 5.180] | 1.765 [0.012 to 3.517] | 2.266 [0.410 to 4.123] | 2.244 [1.155 to 3.333]
  Week 81: number analyzed (Participants) | 10 | 11 | 10 | 31
  Week 81 | 2.153 [-0.046 to 4.352] | 2.422 [-0.327 to 5.170] | 1.971 [-0.291 to 4.233] | 2.190 [0.948 to 3.431]
  Week 89: number analyzed (Participants) | 11 | 10 | 10 | 31
  Week 89 | 2.538 [0.479 to 4.598] | 3.249 [-1.598 to 8.096] | 2.824 [0.109 to 5.539] | 2.860 [1.166 to 4.553]
  Week 97: number analyzed (Participants) | 8 | 11 | 9 | 28
  Week 97 | 1.009 [-0.440 to 2.458] | 2.418 [0.299 to 4.537] | 1.933 [0.279 to 3.587] | 1.860 [0.896 to 2.823]
  Week 110: number analyzed (Participants) | 6 | 11 | 9 | 26
  Week 110 | 0.792 [-0.611 to 2.194] | 3.753 [1.266 to 6.239] | 2.884 [-0.807 to 6.576] | 2.769 [1.226 to 4.311]
  Week 122: number analyzed (Participants) | 4 | 8 | 6 | 18
  Week 122 | -0.133 [-2.124 to 1.859] | 4.543 [1.277 to 7.808] | 1.750 [-0.120 to 3.620] | 2.573 [0.903 to 4.243]
  Week 146: number analyzed (Participants) | 1 | 4 | 4 | 9
  Week 146 | -0.400 [NA to NA] — 95% Confidence Interval was not applicable for individual value. | 5.295 [-5.207 to 15.797] | 4.978 [-1.086 to 11.041] | 4.521 [0.662 to 8.381]
  Week 170: number analyzed (Participants) | 0 | 1 | 1 | 2
  Week 170 |  | 13.780 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 4.300 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 9.040 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval.

37. Secondary Outcome: Change From Baseline on the NSAA - Time to Complete 10 m Run/Walk - B5161004 Baseline
Description: A time to event analysis was performed for loss of ambulation. Loss of ambulation was defined as the inability to walk unassisted and without braces for at least 10 m, as assessed and reported by the investigator at each study visit, and confirmed by the inability to walk/run 10 m (as 1 component of the NSAA) evaluated at the next visit at which timed function tests were performed.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49, 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Seconds
  Baseline: number analyzed (Participants) | 11 | 12 | 9 | 32
  Baseline | 6.245 [4.910 to 7.579] | 5.894 [4.694 to 7.094] | 5.800 [4.789 to 6.811] | 5.988 [5.361 to 6.615]
  Week 13: number analyzed (Participants) | 11 | 12 | 9 | 32
  Week 13 | -0.029 [-0.310 to 0.252] | 0.383 [-1.262 to 2.027] | 0.089 [-0.195 to 0.372] | 0.158 [-0.412 to 0.729]
  Week 25: number analyzed (Participants) | 8 | 9 | 7 | 24
  Week 25 | 0.546 [-0.235 to 1.328] | -0.172 [-1.410 to 1.066] | 0.743 [-0.231 to 1.717] | 0.334 [-0.204 to 0.872]
  Week 49: number analyzed (Participants) | 4 | 4 | 4 | 12
  Week 49 | 0.665 [-0.546 to 1.864] | -0.735 [-4.419 to 2.949] | 0.488 [-0.822 to 1.797] | 0.139 [-0.809 to 1.087]
  Week 73: number analyzed (Participants) | 1 | 2 | 1 | 4
  Week 73 | 1.160 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.480 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.600 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.680 [-0.389 to 1.749]

38. Secondary Outcome: Change From Baseline on the NSAA - Time to Complete 10 m Run/Walk - Overall Baseline
Description: A time to event analysis was performed for loss of ambulation. Loss of ambulation was defined as the inability to walk unassisted and without braces for at least 10 m, as assessed and reported by the investigator at each study visit, and confirmed by the inability to walk/run 10 m (as 1 component of the NSAA) evaluated at the next visit at which timed function tests were performed. This is the overall change from baseline which included the change since enrolling in the parent study B5161002.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was counted starting from the study treatment in study B5161002.
Time Frame: Baseline, Weeks 9,17,25,33,41,49,57,65,73,81,89,97,110,122,146,170.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Seconds
  Baseline: number analyzed (Participants) | 19 | 18 | 18 | 55
  Baseline | 5.780 [5.031 to 6.529] | 5.862 [5.073 to 6.652] | 6.609 [5.596 to 7.623] | 6.078 [5.606 to 6.550]
  Week 9: number analyzed (Participants) | 19 | 17 | 16 | 52
  Week 9 | 0.159 [-0.111 to 0.430] | 0.008 [-0.235 to 0.251] | 0.114 [-0.460 to 0.689] | 0.096 [-0.106 to 0.298]
  Week 17: number analyzed (Participants) | 17 | 15 | 15 | 47
  Week 17 | 0.173 [-0.154 to 0.500] | 0.115 [-0.268 to 0.497] | 0.083 [-0.610 to 0.776] | 0.126 [-0.131 to 0.382]
  Week 25: number analyzed (Participants) | 19 | 17 | 15 | 51
  Week 25 | 0.468 [0.182 to 0.754] | 0.719 [-0.192 to 1.631] | 0.110 [-0.480 to 0.700] | 0.446 [0.101 to 0.792]
  Week 33: number analyzed (Participants) | 19 | 17 | 14 | 50
  Week 33 | 0.348 [-0.109 to 0.805] | 0.417 [-0.241 to 1.076] | 0.264 [-0.319 to 0.846] | 0.348 [0.044 to 0.651]
  Week 41: number analyzed (Participants) | 17 | 16 | 13 | 46
  Week 41 | 0.445 [-0.040 to 0.930] | 0.471 [-0.314 to 1.256] | 0.845 [-0.091 to 1.782] | 0.567 [0.179 to 0.956]
  Week 49: number analyzed (Participants) | 15 | 16 | 13 | 44
  Week 49 | 0.360 [-0.117 to 0.837] | 0.869 [-0.326 to 2.065] | 0.145 [-0.655 to 0.945] | 0.482 [-0.007 to 0.970]
  Week 57: number analyzed (Participants) | 16 | 16 | 11 | 43
  Week 57 | 1.018 [0.383 to 1.653] | 1.573 [-0.263 to 3.408] | 0.539 [-0.214 to 1.292] | 1.102 [0.399 to 1.804]
  Week 65: number analyzed (Participants) | 18 | 15 | 12 | 45
  Week 65 | 1.482 [0.572 to 2.391] | 0.988 [0.190 to 1.786] | 0.745 [-0.069 to 1.559] | 1.121 [0.649 to 1.592]
  Week 73: number analyzed (Participants) | 17 | 15 | 11 | 43
  Week 73 | 1.156 [0.242 to 2.071] | 1.128 [-0.014 to 2.270] | 0.324 [-0.494 to 1.142] | 0.933 [0.391 to 1.476]
  Week 81: number analyzed (Participants) | 15 | 12 | 12 | 39
  Week 81 | 1.243 [0.311 to 2.174] | 0.625 [-0.033 to 1.283] | 0.687 [-0.406 to 1.779] | 0.882 [0.391 to 1.372]
  Week 89: number analyzed (Participants) | 14 | 11 | 11 | 36
  Week 89 | 1.287 [0.332 to 2.242] | 0.837 [0.102 to 1.572] | 0.460 [-0.469 to 1.389] | 0.897 [0.415 to 1.379]
  Week 97: number analyzed (Participants) | 14 | 12 | 11 | 37
  Week 97 | 0.928 [0.193 to 1.663] | 0.883 [-0.405 to 2.172] | 0.670 [-0.393 to 1.733] | 0.837 [0.304 to 1.369]
  Week 110: number analyzed (Participants) | 12 | 13 | 9 | 34
  Week 110 | 1.085 [0.048 to 2.122] | 1.238 [0.382 to 2.095] | 0.300 [-0.800 to 1.400] | 0.936 [0.410 to 1.462]
  Week 122: number analyzed (Participants) | 8 | 10 | 7 | 25
  Week 122 | 1.195 [-0.064 to 2.454] | 1.416 [0.650 to 2.182] | 0.914 [-0.008 to 1.837] | 1.205 [0.719 to 1.690]
  Week 146: number analyzed (Participants) | 4 | 4 | 5 | 13
  Week 146 | 2.138 [-0.866 to 5.141] | 1.588 [-1.542 to 4.717] | 1.662 [0.096 to 3.228] | 1.785 [0.840 to 2.731]
  Week 170: number analyzed (Participants) | 1 | 2 | 1 | 4
  Week 170 | 3.300 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 2.090 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 1.800 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 2.320 [-1.110 to 5.750]

39. Secondary Outcome: Change From Baseline on the Ankle Range of Motion (ROM) - B5161004 Baseline
Description: ROM of the ankle was evaluated by goniometry and any occurrences of ankle contractures were recorded. In order to provide optimal testing conditions and consistency in endpoint measurements, the functional assessment of ankle ROM was completed at approximately the same time of day.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49 and 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Degrees of Passive Flexion
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Degrees of Passive Flexion
  Left Ankle - Baseline: number analyzed (Participants) | 16 | 16 | 18 | 50
  Left Ankle - Baseline | 0.6 [-3.7 to 4.8] | -0.4 [-6.8 to 5.9] | -7.8 [-13.8 to -1.9] | -2.8 [-6.0 to 0.4]
  Left Ankle - Week 13: number analyzed (Participants) | 16 | 16 | 17 | 49
  Left Ankle - Week 13 | -2.1 [-5.2 to 1.0] | -1.0 [-5.2 to 3.2] | -0.9 [-3.7 to 1.8] | -1.3 [-3.2 to 0.5]
  Left Ankle - Week 25: number analyzed (Participants) | 11 | 12 | 14 | 37
  Left Ankle - Week 25 | -2.2 [-5.4 to 1.0] | -1.8 [-8.7 to 5.0] | -2.4 [-6.4 to 1.5] | -2.2 [-4.7 to 0.4]
  Left Ankle - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Left Ankle - Week 49 | -1.7 [-12.0 to 8.6] | -6.2 [-15.2 to 2.9] | -4.0 [-11.4 to 3.4] | -3.9 [-8.1 to 0.4]
  Left Ankle - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Left Ankle - Week 73 | -2.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -3.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.7 [-6.8 to 3.4]
  Right Ankle - Baseline: number analyzed (Participants) | 16 | 16 | 18 | 50
  Right Ankle - Baseline | 0.0 [-4.2 to 4.2] | -3.1 [-10.3 to 4.2] | -10.3 [-17.9 to -2.7] | -4.7 [-8.5 to -0.9]
  Right Ankle - Week 13: number analyzed (Participants) | 16 | 16 | 17 | 49
  Right Ankle - Week 13 | -0.8 [-4.5 to 3.0] | 0.4 [-3.0 to 3.9] | 0.8 [-2.1 to 3.7] | 0.2 [-1.6 to 2.0]
  Right Ankle - Week 25: number analyzed (Participants) | 11 | 12 | 14 | 37
  Right Ankle - Week 25 | -1.5 [-5.3 to 2.2] | -1.7 [-7.0 to 3.6] | -2.1 [-6.0 to 1.8] | -1.8 [-4.1 to 0.5]
  Right Ankle - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Right Ankle - Week 49 | -4.1 [-12.3 to 4.0] | -3.3 [-6.1 to -0.5] | -3.0 [-6.1 to 0.1] | -3.5 [-6.1 to -0.9]
  Right Ankle - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Right Ankle - Week 73 | -1.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 3.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 5.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 2.5 [-7.1 to 12.1]

40. Secondary Outcome: Change From Baseline on the Ankle ROM - Overall Baseline
Description: ROM of the ankle was evaluated by goniometry and any occurrences of ankle contractures were recorded. In order to provide optimal testing conditions and consistency in endpoint measurements, the functional assessment of ankle ROM was completed at approximately the same time of day. This is the overall change from baseline which included the change since enrolling in the parent study B5161002.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was counted starting from the study treatment in study B5161002.
Time Frame: Baseline, Weeks 9,17,25,33,41,49,57,65,73,81,89,97,110,122,146,170.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Degrees of Passive Flexion
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Degrees of Passive Flexion
  Left Ankle - Baseline | 7.1 [4.7 to 9.5] | 2.6 [-1.8 to 6.9] | 1.6 [-1.3 to 4.4] | 3.7 [1.8 to 5.6]
  Left Ankle - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Left Ankle - Week 9 | -1.8 [-4.1 to 0.4] | -0.8 [-3.6 to 2.1] | -0.2 [-2.7 to 2.3] | -0.9 [-2.3 to 0.5]
  Left Ankle - Week 17 | -2.5 [-5.5 to 0.4] | -2.0 [-4.4 to 0.4] | -1.0 [-3.4 to 1.4] | -1.8 [-3.2 to -0.4]
  Left Ankle - Week 25: number analyzed (Participants) | 19 | 20 | 19 | 58
  Left Ankle - Week 25 | -2.3 [-5.5 to 1.0] | -4.7 [-7.6 to -1.8] | 0.0 [-2.0 to 2.0] | -2.4 [-3.9 to -0.8]
  Left Ankle - Week 33 | -1.1 [-4.9 to 2.7] | -2.4 [-5.1 to 0.3] | -1.9 [-3.8 to 0.0] | -1.8 [-3.4 to -0.2]
  Left Ankle - Week 41: number analyzed (Participants) | 18 | 20 | 20 | 58
  Left Ankle - Week 41 | -2.4 [-6.0 to 1.2] | -3.8 [-6.3 to -1.2] | -2.1 [-4.6 to 0.4] | -2.8 [-4.3 to -1.2]
  Left Ankle - Week 49 | -3.2 [-6.6 to 0.2] | -5.5 [-8.9 to -2.1] | -2.3 [-5.4 to 0.9] | -3.7 [-5.5 to -1.8]
  Left Ankle - Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Left Ankle - Week 57 | -3.5 [-6.5 to -0.6] | -6.1 [-10.4 to -1.7] | -5.8 [-10.0 to -1.6] | -5.1 [-7.3 to -3.0]
  Left Ankle - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Left Ankle - Week 65 | -4.1 [-7.8 to -0.3] | -5.4 [-12.6 to 1.9] | -5.2 [-9.3 to -1.1] | -4.9 [-7.8 to -2.0]
  Left Ankle - Week 73 | -2.5 [-6.6 to 1.6] | -4.6 [-12.2 to 3.1] | -6.6 [-10.4 to -2.7] | -4.6 [-7.6 to -1.5]
  Left Ankle - Week 81: number analyzed (Participants) | 19 | 18 | 20 | 57
  Left Ankle - Week 81 | -6.1 [-10.7 to -1.5] | -2.7 [-9.6 to 4.3] | -8.7 [-13.2 to -4.1] | -5.9 [-8.9 to -2.9]
  Left Ankle - Week 89: number analyzed (Participants) | 18 | 20 | 19 | 57
  Left Ankle - Week 89 | -9.9 [-16.2 to -3.7] | -6.3 [-16.0 to 3.4] | -8.4 [-13.6 to -3.1] | -8.1 [-12.2 to -4.1]
  Left Ankle - Week 97 | -7.9 [-14.1 to -1.8] | -10.0 [-16.7 to -3.2] | -9.3 [-13.7 to -4.8] | -9.1 [-12.2 to -5.9]
  Left Ankle - Week 110: number analyzed (Participants) | 16 | 16 | 17 | 49
  Left Ankle - Week 110 | -8.3 [-14.2 to -2.4] | -5.9 [-12.8 to 1.0] | -9.9 [-15.4 to -4.4] | -8.1 [-11.4 to -4.8]
  Left Ankle - Week 122: number analyzed (Participants) | 11 | 12 | 14 | 37
  Left Ankle - Week 122 | -8.7 [-16.4 to -1.1] | -5.7 [-12.8 to 1.5] | -11.5 [-19.0 to -4.0] | -8.8 [-12.7 to -4.8]
  Left Ankle - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Left Ankle - Week 146 | -10.0 [-21.7 to 1.7] | -10.8 [-19.7 to -1.9] | -10.9 [-22.9 to 1.2] | -10.6 [-15.7 to -5.4]
  Left Ankle - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Left Ankle - Week 170 | -6.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -6.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -9.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -7.2 [-13.4 to -1.0]
  Right Ankle - Baseline | 6.7 [4.4 to 9.1] | 1.0 [-4.0 to 6.0] | 1.5 [-1.6 to 4.6] | 3.0 [0.9 to 5.1]
  Right Ankle - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Right Ankle - Week 9 | -1.9 [-5.0 to 1.2] | -0.8 [-3.5 to 1.9] | -1.3 [-3.6 to 1.0] | -1.3 [-2.8 to 0.2]
  Right Ankle - Week 17 | -2.2 [-6.3 to 2.0] | -1.8 [-3.9 to 0.3] | -2.0 [-4.8 to 0.9] | -2.0 [-3.7 to -0.3]
  Right Ankle - Week 25 | -1.5 [-5.2 to 2.1] | -4.5 [-7.6 to -1.3] | -3.1 [-5.8 to -0.4] | -3.1 [-4.8 to -1.3]
  Right Ankle - Week 33 | 0.4 [-3.7 to 4.5] | -1.6 [-4.7 to 1.6] | -3.4 [-5.9 to -0.8] | -1.5 [-3.3 to 0.3]
  Right Ankle - Week 41 | -2.7 [-6.0 to 0.6] | -3.1 [-6.0 to -0.1] | -2.7 [-5.7 to 0.4] | -2.8 [-4.5 to -1.1]
  Right Ankle - Week 49 | -3.8 [-7.6 to -0.1] | -4.5 [-7.9 to -1.1] | -2.5 [-6.3 to 1.4] | -3.6 [-5.6 to -1.6]
  Right Ankle - Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Right Ankle - Week 57 | -2.5 [-6.1 to 1.0] | -5.3 [-9.8 to -0.8] | -7.9 [-12.4 to -3.5] | -5.2 [-7.6 to -2.9]
  Right Ankle - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Right Ankle - Week 65 | -4.7 [-9.1 to -0.4] | -5.4 [-12.6 to 1.9] | -6.6 [-10.8 to -2.4] | -5.6 [-8.5 to -2.6]
  Right Ankle - Week 73 | -3.6 [-8.0 to 0.8] | -3.0 [-10.1 to 4.2] | -8.0 [-12.6 to -3.4] | -4.9 [-7.9 to -1.8]
  Right Ankle - Week 81: number analyzed (Participants) | 19 | 18 | 20 | 57
  Right Ankle - Week 81 | -5.1 [-9.7 to -0.5] | -1.4 [-7.9 to 5.1] | -10.0 [-14.9 to -5.1] | -5.6 [-8.7 to -2.6]
  Right Ankle - Week 89: number analyzed (Participants) | 18 | 20 | 19 | 57
  Right Ankle - Week 89 | -9.4 [-15.4 to -3.4] | -6.8 [-15.4 to 1.9] | -10.4 [-15.8 to -5.0] | -8.8 [-12.6 to -5.0]
  Right Ankle - Week 97 | -7.5 [-12.4 to -2.5] | -10.6 [-18.3 to -2.9] | -11.8 [-17.5 to -6.1] | -10.0 [-13.4 to -6.6]
  Right Ankle - Week 110: number analyzed (Participants) | 16 | 16 | 17 | 49
  Right Ankle - Week 110 | -7.4 [-13.9 to -0.9] | -5.9 [-11.6 to -0.2] | -10.4 [-16.4 to -4.3] | -7.9 [-11.2 to -4.6]
  Right Ankle - Week 122: number analyzed (Participants) | 11 | 12 | 14 | 37
  Right Ankle - Week 122 | -7.6 [-14.9 to -0.3] | -6.8 [-14.3 to 0.6] | -12.7 [-20.1 to -5.3] | -9.3 [-13.3 to -5.3]
  Right Ankle - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Right Ankle - Week 146 | -12.6 [-24.4 to -0.7] | -9.2 [-20.6 to 2.2] | -12.1 [-23.5 to -0.7] | -11.4 [-16.8 to -6.0]
  Right Ankle - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Right Ankle - Week 170 | -7.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -3.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -12.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -7.7 [-16.3 to 1.0]

41. Secondary Outcome: Change From Baseline on the Performance of Upper Limb (PUL) Overall Score - B5161004 Baseline
Description: The PUL scale was used to assess motor performance of the upper limb for individuals with DMD. The PUL scale includes 22 items; an entry item defining the starting functional level, and 21 items subdivided into 3 levels; shoulder (4 items), middle (9 items) and distal (8 items). Scoring options per item may not be uniform and may vary from 0-1 to 0-6, according to the performance, with higher values corresponding to better performance. A total maximum score of 74 is achieved by adding the individual level scores; shoulder maximum 16, middle level maximum score 34 and distal level maximum score 24. In order to provide optimal testing conditions and consistency in endpoint measurements, the functional assessment of PUL was completed at approximately the same time of day.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49 and 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Units on a Scale
  Baseline: number analyzed (Participants) | 15 | 16 | 17 | 48
  Baseline | 65.6 [63.0 to 68.2] | 65.3 [61.4 to 69.1] | 63.8 [59.9 to 67.8] | 64.9 [62.9 to 66.8]
  Week 13: number analyzed (Participants) | 14 | 16 | 16 | 46
  Week 13 | -1.2 [-2.3 to -0.1] | -1.5 [-2.6 to -0.4] | -1.8 [-3.7 to 0.0] | -1.5 [-2.3 to -0.8]
  Week 25: number analyzed (Participants) | 9 | 11 | 13 | 33
  Week 25 | -1.2 [-2.3 to -0.2] | -3.0 [-5.3 to -0.7] | -0.3 [-1.2 to 0.6] | -1.5 [-2.4 to -0.6]
  Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Week 49 | -1.6 [-5.5 to 2.4] | -7.8 [-14.1 to -1.6] | -2.6 [-6.3 to 1.1] | -3.8 [-6.3 to -1.3]
  Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Week 73 | -13.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -7.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -6.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -9.0 [-15.0 to -3.0]

42. Secondary Outcome: Change From Baseline on the PUL Overall Score - Overall Baseline
Description: The PUL scale was used to assess motor performance of the upper limb for individuals with DMD. The PUL scale includes 22 items; an entry item defining the starting functional level, and 21 items subdivided into 3 levels; shoulder (4 items), middle (9 items) and distal (8 items). Scoring options per item may not be uniform and may vary from 0-1 to 0-6, according to the performance, with higher values corresponding to better performance. A total maximum score of 74 is achieved by adding the individual level scores; shoulder maximum 16, middle level maximum score 34 and distal level maximum score 24.
  This is the overall change from baseline which included the change since enrolling in parent study B5161002. Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was counted starting from the study treatment in study B5161002.
Time Frame: Baseline, Weeks 9,17,25,33,41,49,57,65,73,81,89,97,110,122,146,170.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Units on a Scale
  Baseline | 66.3 [65.0 to 67.6] | 66.9 [64.7 to 69.0] | 66.9 [65.1 to 68.6] | 66.7 [65.7 to 67.6]
  Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Week 9 | -0.7 [-2.0 to 0.5] | 0.5 [-0.7 to 1.7] | -0.1 [-1.0 to 0.8] | -0.1 [-0.7 to 0.5]
  Week 17: number analyzed (Participants) | 19 | 20 | 19 | 58
  Week 17 | -0.5 [-2.6 to 1.5] | -0.2 [-1.3 to 0.9] | -0.4 [-3.1 to 2.2] | -0.4 [-1.5 to 0.7]
  Week 25: number analyzed (Participants) | 18 | 19 | 20 | 57
  Week 25 | 0.7 [-1.1 to 2.4] | 0.3 [-0.6 to 1.1] | 0.2 [-1.5 to 1.8] | 0.4 [-0.5 to 1.2]
  Week 33 | 0.5 [-0.8 to 1.9] | -0.5 [-2.4 to 1.4] | -0.5 [-1.7 to 0.7] | -0.2 [-1.0 to 0.7]
  Week 41: number analyzed (Participants) | 18 | 20 | 20 | 58
  Week 41 | -0.1 [-2.1 to 2.0] | -0.4 [-1.9 to 1.2] | -0.4 [-1.9 to 1.2] | -0.3 [-1.2 to 0.7]
  Week 49 | 0.1 [-1.6 to 1.8] | -0.8 [-2.9 to 1.4] | -0.5 [-1.9 to 0.9] | -0.4 [-1.4 to 0.6]
  Week 57: number analyzed (Participants) | 19 | 17 | 19 | 55
  Week 57 | -0.3 [-2.2 to 1.5] | -0.8 [-2.9 to 1.4] | -4.7 [-12.0 to 2.6] | -2.0 [-4.6 to 0.6]
  Week 65: number analyzed (Participants) | 18 | 20 | 20 | 58
  Week 65 | 0.6 [-1.0 to 2.2] | -0.9 [-3.0 to 1.3] | -4.6 [-11.6 to 2.5] | -1.7 [-4.2 to 0.8]
  Week 73 | -1.0 [-2.9 to 0.9] | -1.8 [-4.5 to 0.9] | -1.2 [-3.3 to 1.0] | -1.3 [-2.6 to -0.1]
  Week 81: number analyzed (Participants) | 19 | 19 | 19 | 57
  Week 81 | -0.7 [-2.5 to 1.1] | -1.2 [-3.7 to 1.4] | -1.5 [-3.7 to 0.6] | -1.1 [-2.3 to 0.1]
  Week 89: number analyzed (Participants) | 18 | 20 | 20 | 58
  Week 89 | -0.4 [-2.0 to 1.1] | -2.9 [-7.0 to 1.2] | -2.3 [-4.5 to -0.1] | -1.9 [-3.5 to -0.3]
  Week 97: number analyzed (Participants) | 18 | 19 | 19 | 56
  Week 97 | -1.4 [-3.9 to 1.0] | -2.2 [-5.3 to 0.9] | -2.3 [-5.1 to 0.4] | -2.0 [-3.5 to -0.5]
  Week 110: number analyzed (Participants) | 15 | 17 | 17 | 49
  Week 110 | -1.5 [-3.7 to 0.7] | -3.2 [-6.7 to 0.2] | -4.4 [-8.5 to -0.4] | -3.1 [-5.0 to -1.3]
  Week 122: number analyzed (Participants) | 10 | 12 | 13 | 35
  Week 122 | -1.4 [-5.3 to 2.5] | -2.8 [-6.8 to 1.3] | -2.4 [-5.4 to 0.6] | -2.2 [-4.1 to -0.3]
  Week 146: number analyzed (Participants) | 7 | 6 | 8 | 21
  Week 146 | -2.3 [-7.4 to 2.9] | -6.8 [-15.3 to 1.6] | -2.9 [-7.7 to 2.0] | -3.8 [-6.7 to -0.9]
  Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Week 170 | -14.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -4.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -9.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -9.0 [-17.8 to -0.2]

43. Secondary Outcome: Change From Baseline on the Six Minute Walk Distance (6MWD) - B5161004 Baseline
Description: The 6MWD evaluated ambulation ability by measuring the distance walked in 6 minutes. In order to provide optimal testing conditions and consistency in endpoint measurements, the functional assessment of 6MWD was completed at approximately the same time of day.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49 and 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Meters
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Meters
  Baseline: number analyzed (Participants) | 15 | 13 | 11 | 39
  Baseline | 328.0 [266.5 to 389.5] | 386.2 [341.1 to 431.2] | 360.4 [305.1 to 415.6] | 356.5 [326.3 to 386.8]
  Week 13: number analyzed (Participants) | 15 | 13 | 11 | 39
  Week 13 | -23.6 [-50.0 to 2.8] | -26.1 [-45.6 to -6.5] | -8.4 [-28.6 to 11.9] | -20.1 [-32.5 to -7.7]
  Week 25: number analyzed (Participants) | 10 | 10 | 8 | 28
  Week 25 | -45.5 [-83.4 to -7.6] | -16.1 [-37.4 to 5.2] | -11.3 [-37.6 to 15.1] | -25.2 [-41.3 to -9.1]
  Week 49: number analyzed (Participants) | 6 | 5 | 6 | 17
  Week 49 | -98.0 [-219.5 to 23.5] | -16.8 [-55.2 to 21.6] | -39.0 [-68.2 to -9.8] | -53.3 [-92.8 to -13.8]
  Week 73: number analyzed (Participants) | 2 | 2 | 1 | 5
  Week 73 | -110.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -41.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -22.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -65.0 [-124.4 to -5.6]

44. Secondary Outcome: Change From Baseline on the 6MWD - Overall Baseline
Description: The 6MWD evaluated ambulation ability by measuring the distance walked in 6 minutes. In order to provide optimal testing conditions and consistency in endpoint measurements, the functional assessment of 6MWD was completed at approximately the same time of day. This is the overall change from baseline which included the change since enrolling in the parent study B5161002.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was start of the study treatment in parent study B5161002.
Time Frame: Baseline,Weeks 9,17,25,33,41,49,57,65,73,81,89,97,110,122,146,170.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Meters
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Meters
  Baseline | 409.1 [367.2 to 450.9] | 349.4 [290.3 to 408.5] | 363.7 [326.0 to 401.4] | 373.5 [347.0 to 399.9]
  Week 9: number analyzed (Participants) | 18 | 17 | 19 | 54
  Week 9 | -11.6 [-29.5 to 6.3] | -2.0 [-22.8 to 18.8] | -9.3 [-21.3 to 2.7] | -7.8 [-17.0 to 1.4]
  Week 17: number analyzed (Participants) | 19 | 17 | 18 | 54
  Week 17 | -36.8 [-63.9 to -9.7] | -16.1 [-39.2 to 7.1] | -15.6 [-34.8 to 3.6] | -23.2 [-36.2 to -10.2]
  Week 25: number analyzed (Participants) | 17 | 18 | 17 | 52
  Week 25 | -41.8 [-80.7 to -2.9] | -8.2 [-35.7 to 19.3] | -29.6 [-54.9 to -4.4] | -26.2 [-43.3 to -9.1]
  Week 33: number analyzed (Participants) | 19 | 18 | 17 | 54
  Week 33 | -43.8 [-74.2 to -13.5] | -17.5 [-45.8 to 10.8] | -34.9 [-62.3 to -7.5] | -32.3 [-48.1 to -16.4]
  Week 41: number analyzed (Participants) | 17 | 18 | 15 | 50
  Week 41 | -54.2 [-91.3 to -17.1] | -37.4 [-70.8 to -4.1] | -34.9 [-64.2 to -5.7] | -42.4 [-60.6 to -24.1]
  Week 49: number analyzed (Participants) | 18 | 17 | 15 | 50
  Week 49 | -59.8 [-96.8 to -22.9] | -29.1 [-64.2 to 6.0] | -37.3 [-65.9 to -8.8] | -42.6 [-61.4 to -23.8]
  Week 57: number analyzed (Participants) | 18 | 16 | 13 | 47
  Week 57 | -72.2 [-109.9 to -34.4] | -32.8 [-69.8 to 4.1] | -52.6 [-86.8 to -18.4] | -53.4 [-73.7 to -33.0]
  Week 65: number analyzed (Participants) | 17 | 15 | 13 | 45
  Week 65 | -74.5 [-128.9 to -20.0] | -33.3 [-71.1 to 4.5] | -58.2 [-106.3 to -10.0] | -56.0 [-82.2 to -29.8]
  Week 73: number analyzed (Participants) | 17 | 15 | 15 | 47
  Week 73 | -77.2 [-119.8 to -34.7] | -35.5 [-70.6 to -0.4] | -60.1 [-102.5 to -17.6] | -58.4 [-80.6 to -36.3]
  Week 81: number analyzed (Participants) | 17 | 14 | 14 | 45
  Week 81 | -78.9 [-120.5 to -37.3] | -42.6 [-94.7 to 9.5] | -39.6 [-64.4 to -14.7] | -55.4 [-78.0 to -32.7]
  Week 89: number analyzed (Participants) | 16 | 13 | 12 | 41
  Week 89 | -96.7 [-141.5 to -51.9] | -33.7 [-73.3 to 5.9] | -41.5 [-63.8 to -19.2] | -60.6 [-83.2 to -37.9]
  Week 97: number analyzed (Participants) | 17 | 13 | 13 | 43
  Week 97 | -80.7 [-131.4 to -30.1] | -25.1 [-64.0 to 13.9] | -55.3 [-79.3 to -31.3] | -56.2 [-79.8 to -32.6]
  Week 110: number analyzed (Participants) | 16 | 17 | 16 | 49
  Week 110 | -115.5 [-171.8 to -59.2] | -87.9 [-141.6 to -34.1] | -126.1 [-189.2 to -63.0] | -109.4 [-140.6 to -78.2]
  Week 122: number analyzed (Participants) | 11 | 12 | 13 | 36
  Week 122 | -142.5 [-229.0 to -56.1] | -69.8 [-144.7 to 5.0] | -155.0 [-231.0 to -79.0] | -122.8 [-165.6 to -80.0]
  Week 146: number analyzed (Participants) | 6 | 6 | 7 | 19
  Week 146 | -224.0 [-454.5 to 6.5] | -53.2 [-179.5 to 73.2] | -137.1 [-209.0 to -65.3] | -138.1 [-213.2 to -62.9]
  Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Week 170 | -184.0 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -90.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -206.5 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -160.3 [-294.3 to -26.4]

45. Secondary Outcome: Change From Baseline on the Forced Expiratory Volume in One Second (FEV1) - B5161004 Baseline
Description: The FEV1 was recorded as an absolute volume in litres and in terms of predicted values according to age, height, race and gender. The best single FEV1 measurement from a set of 3 was recorded in the database.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49 and 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Litres
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Litres
  FEV1 - Baseline: number analyzed (Participants) | 16 | 17 | 17 | 50
  FEV1 - Baseline | 1.3694 [1.1372 to 1.6015] | 1.4235 [1.1693 to 1.6777] | 1.5335 [1.3687 to 1.6983] | 1.4436 [1.3243 to 1.5629]
  FEV1 - Week 13: number analyzed (Participants) | 16 | 15 | 14 | 45
  FEV1 - Week 13 | 0.1113 [-0.0094 to 0.2319] | 0.1307 [-0.0040 to 0.2653] | -0.0014 [-0.1178 to 0.1150] | 0.0827 [0.0144 to 0.1509]
  FEV1 - Week 25: number analyzed (Participants) | 11 | 12 | 13 | 36
  FEV1 - Week 25 | 0.1473 [-0.0405 to 0.3351] | 0.1175 [0.0093 to 0.2257] | 0.0923 [-0.0524 to 0.2370] | 0.1175 [0.0406 to 0.1944]
  FEV1 - Week 49: number analyzed (Participants) | 7 | 6 | 6 | 19
  FEV1 - Week 49 | 0.3057 [0.0016 to 0.6098] | 0.2083 [-0.0561 to 0.4728] | 0.1000 [-0.0167 to 0.2167] | 0.2100 [0.0874 to 0.3326]
  FEV1 - Week 73: number analyzed (Participants) | 2 | 2 | 1 | 5
  FEV1 - Week 73 | 0.7500 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.2550 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.2800 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.4580 [-0.3052 to 1.2212]

46. Secondary Outcome: Change From Baseline on the Peak Expiratory Flow Rate (PEFR)- B5161004 Baseline
Description: PEFR was one of the Pulmonary Function Tests (PFTs). Three technically adequate peak expiratory flow rate (PEFR) maneuvers were performed and reported in Litres/Minute (L/min), and the highest single PEFR was reported in the database. In order to provide optimal testing conditions and consistency in endpoint measurements, the functional assessment of PEFR was completed at approximately the same time of day.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49 and 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: L/min
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
L/min
  Baseline: number analyzed (Participants) | 14 | 17 | 17 | 48
  Baseline | 200.314 [154.281 to 246.348] | 187.200 [150.135 to 224.265] | 185.882 [163.694 to 208.071] | 190.558 [171.737 to 209.380]
  Week 13: number analyzed (Participants) | 14 | 15 | 14 | 43
  Week 13 | -17.014 [-56.536 to 22.507] | 20.613 [-8.846 to 50.073] | 8.214 [-29.197 to 45.626] | 4.326 [-15.003 to 23.654]
  Week 25: number analyzed (Participants) | 10 | 12 | 12 | 34
  Week 25 | -16.260 [-59.079 to 26.559] | 0.767 [-22.311 to 23.845] | 39.250 [6.034 to 72.466] | 9.341 [-9.379 to 28.061]
  Week 49: number analyzed (Participants) | 7 | 6 | 6 | 19
  Week 49 | -31.171 [-94.943 to 32.600] | 11.700 [-55.267 to 78.667] | 50.967 [-1.595 to 103.529] | 8.305 [-24.489 to 41.099]
  Week 73: number analyzed (Participants) | 2 | 2 | 1 | 5
  Week 73 | 6.800 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 5.600 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 36.000 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 12.160 [-81.893 to 106.213]

47. Secondary Outcome: Change From Baseline on the Myometry Based Muscle Strength - B5161004 Baseline
Description: Muscle strength was quantified by means of a handheld dynamometer. The following muscle groups were evaluated: knee extension, elbow flexion, elbow extension, hip abduction and shoulder abduction. 95% Confidence Interval was not calculated when less than or equal to 3 participants' data were available.
  Baseline was defined as the last assessment prior to dosing on Day 1 in B5161004. Week 1 was counted starting from the study treatment in study B5161004.
Time Frame: Baseline, Weeks 13, 25, 49, 73.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Kilograms
  Elbow Extension-Left - Baseline: number analyzed (Participants) | 16 | 17 | 18 | 51
  Elbow Extension-Left - Baseline | 3.35 [2.47 to 4.23] | 3.24 [2.58 to 3.89] | 2.83 [2.13 to 3.52] | 3.13 [2.72 to 3.53]
  Elbow Extension-Left - Week 13: number analyzed (Participants) | 16 | 17 | 17 | 50
  Elbow Extension-Left - Week 13 | -0.21 [-0.55 to 0.14] | -0.55 [-1.11 to 0.01] | -0.31 [-0.81 to 0.18] | -0.36 [-0.62 to -0.10]
  Elbow Extension-Left - Week 25: number analyzed (Participants) | 11 | 12 | 14 | 37
  Elbow Extension-Left - Week 25 | -0.44 [-0.94 to 0.07] | -0.38 [-1.13 to 0.36] | -0.09 [-0.63 to 0.45] | -0.29 [-0.61 to 0.03]
  Elbow Extension-Left - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Elbow Extension-Left - Week 49 | -0.66 [-1.93 to 0.61] | -0.47 [-1.05 to 0.12] | -0.23 [-0.67 to 0.22] | -0.45 [-0.86 to -0.04]
  Elbow Extension-Left - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Elbow Extension-Left - Week 73 | -1.15 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.95 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.10 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.73 [-1.46 to 0.00]
  Elbow Extension-Right - Baseline: number analyzed (Participants) | 16 | 17 | 18 | 51
  Elbow Extension-Right - Baseline | 3.31 [2.36 to 4.26] | 3.24 [2.53 to 3.95] | 2.94 [2.29 to 3.60] | 3.16 [2.74 to 3.57]
  Elbow Extension-Right - Week 13: number analyzed (Participants) | 16 | 17 | 17 | 50
  Elbow Extension-Right - Week 13 | -0.23 [-0.61 to 0.15] | -0.42 [-1.05 to 0.21] | -0.27 [-0.71 to 0.17] | -0.31 [-0.58 to -0.04]
  Elbow Extension-Right - Week 25: number analyzed (Participants) | 10 | 12 | 14 | 36
  Elbow Extension-Right - Week 25 | -0.40 [-1.05 to 0.25] | -0.68 [-1.21 to -0.14] | 0.06 [-0.41 to 0.53] | -0.31 [-0.61 to -0.01]
  Elbow Extension-Right - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Elbow Extension-Right - Week 49 | -0.59 [-1.82 to 0.65] | -0.60 [-1.07 to -0.13] | -0.07 [-0.55 to 0.41] | -0.41 [-0.82 to 0.00]
  Elbow Extension-Right - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Elbow Extension-Right - Week 73 | -0.70 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.25 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.20 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.58 [-1.35 to 0.18]
  Elbow Flexion-Left - Baseline: number analyzed (Participants) | 16 | 17 | 18 | 51
  Elbow Flexion-Left - Baseline | 4.14 [2.79 to 5.49] | 3.74 [3.01 to 4.46] | 3.19 [2.50 to 3.88] | 3.67 [3.15 to 4.19]
  Elbow Flexion-Left - Week 13: number analyzed (Participants) | 16 | 17 | 17 | 50
  Elbow Flexion-Left - Week 13 | -0.49 [-1.15 to 0.17] | -0.22 [-0.92 to 0.49] | -0.36 [-0.85 to 0.12] | -0.35 [-0.69 to -0.02]
  Elbow Flexion-Left - Week 25: number analyzed (Participants) | 11 | 12 | 14 | 37
  Elbow Flexion-Left - Week 25 | -0.65 [-1.50 to 0.21] | -0.58 [-1.69 to 0.52] | -0.19 [-0.54 to 0.15] | -0.45 [-0.87 to -0.04]
  Elbow Flexion-Left - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Elbow Flexion-Left - Week 49 | -1.13 [-2.97 to 0.71] | -0.08 [-1.33 to 1.16] | -0.39 [-1.10 to 0.33] | -0.56 [-1.22 to 0.11]
  Elbow Flexion-Left - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Elbow Flexion-Left - Week 73 | -1.25 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.55 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.05 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.95 [-2.09 to 0.19]
  Elbow Flexion - Right - Baseline: number analyzed (Participants) | 16 | 17 | 18 | 51
  Elbow Flexion - Right - Baseline | 4.13 [2.85 to 5.40] | 4.18 [3.33 to 5.02] | 3.07 [2.45 to 3.69] | 3.77 [3.25 to 4.28]
  Elbow Flexion - Right - Week 13: number analyzed (Participants) | 16 | 17 | 17 | 50
  Elbow Flexion - Right - Week 13 | -0.48 [-1.15 to 0.20] | -0.85 [-1.53 to -0.17] | -0.18 [-0.50 to 0.14] | -0.50 [-0.82 to -0.18]
  Elbow Flexion - Right - Week 25: number analyzed (Participants) | 10 | 12 | 14 | 36
  Elbow Flexion - Right - Week 25 | -0.75 [-2.03 to 0.53] | -1.08 [-2.04 to -0.11] | 0.32 [-0.03 to 0.67] | -0.44 [-0.93 to 0.05]
  Elbow Flexion - Right - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Elbow Flexion - Right - Week 49 | -0.49 [-1.89 to 0.92] | -1.27 [-2.25 to -0.29] | -0.36 [-0.62 to -0.10] | -0.68 [-1.18 to -0.17]
  Elbow Flexion - Right - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Elbow Flexion - Right - Week 73 | -1.25 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.20 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.70 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.05 [-1.46 to -0.64]
  Hip Abduction - Left - Baseline: number analyzed (Participants) | 16 | 17 | 17 | 50
  Hip Abduction - Left - Baseline | 4.23 [2.91 to 5.54] | 5.29 [4.32 to 6.25] | 4.92 [4.28 to 5.57] | 4.82 [4.28 to 5.37]
  Hip Abduction - Left - Week 13: number analyzed (Participants) | 16 | 17 | 16 | 49
  Hip Abduction - Left - Week 13 | 0.06 [-0.40 to 0.51] | -0.46 [-1.43 to 0.50] | -0.26 [-1.19 to 0.67] | -0.23 [-0.67 to 0.22]
  Hip Abduction - Left - Week 25: number analyzed (Participants) | 10 | 12 | 13 | 35
  Hip Abduction - Left - Week 25 | -0.08 [-1.38 to 1.22] | -0.75 [-1.63 to 0.13] | -0.11 [-0.78 to 0.56] | -0.32 [-0.81 to 0.17]
  Hip Abduction - Left - Week 49: number analyzed (Participants) | 7 | 5 | 7 | 19
  Hip Abduction - Left - Week 49 | -0.81 [-3.04 to 1.41] | -0.94 [-1.98 to 0.10] | 0.00 [-0.72 to 0.72] | -0.55 [-1.30 to 0.21]
  Hip Abduction - Left - Week 73: number analyzed (Participants) | 2 | 2 | 1 | 5
  Hip Abduction - Left - Week 73 | -0.75 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -2.20 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.30 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.12 [-2.83 to 0.59]
  Hip Abduction - Right - Baseline: number analyzed (Participants) | 16 | 17 | 17 | 50
  Hip Abduction - Right - Baseline | 4.39 [2.80 to 5.98] | 5.55 [4.44 to 6.67] | 4.99 [4.23 to 5.75] | 4.99 [4.34 to 5.64]
  Hip Abduction - Right - Week 13: number analyzed (Participants) | 16 | 17 | 16 | 49
  Hip Abduction - Right - Week 13 | -0.04 [-0.59 to 0.52] | -0.75 [-1.94 to 0.43] | -0.51 [-1.42 to 0.41] | -0.44 [-0.95 to 0.07]
  Hip Abduction - Right - Week 25: number analyzed (Participants) | 10 | 12 | 13 | 35
  Hip Abduction - Right - Week 25 | -0.10 [-1.77 to 1.57] | -0.94 [-2.44 to 0.56] | -0.52 [-1.54 to 0.51] | -0.54 [-1.26 to 0.18]
  Hip Abduction - Right - Week 49: number analyzed (Participants) | 7 | 5 | 7 | 19
  Hip Abduction - Right - Week 49 | -1.10 [-3.88 to 1.68] | -0.66 [-2.74 to 1.42] | 0.01 [-1.33 to 1.36] | -0.57 [-1.61 to 0.46]
  Hip Abduction - Right - Week 73: number analyzed (Participants) | 2 | 2 | 1 | 5
  Hip Abduction - Right - Week 73 | -0.30 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -2.15 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.30 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.92 [-3.05 to 1.21]
  Knee Extension - Left - Baseline: number analyzed (Participants) | 16 | 17 | 18 | 51
  Knee Extension - Left - Baseline | 4.21 [3.01 to 5.40] | 4.54 [3.40 to 5.68] | 4.59 [3.10 to 6.08] | 4.45 [3.76 to 5.15]
  Knee Extension - Left - Week 13: number analyzed (Participants) | 16 | 17 | 17 | 50
  Knee Extension - Left - Week 13 | -0.34 [-0.99 to 0.30] | -0.44 [-1.28 to 0.40] | -1.02 [-1.85 to -0.19] | -0.61 [-1.04 to -0.18]
  Knee Extension - Left - Week 25: number analyzed (Participants) | 11 | 12 | 14 | 37
  Knee Extension - Left - Week 25 | -0.60 [-1.37 to 0.17] | -0.73 [-1.85 to 0.38] | -0.92 [-1.66 to -0.18] | -0.76 [-1.23 to -0.30]
  Knee Extension - Left - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Knee Extension - Left - Week 49 | -0.34 [-1.15 to 0.46] | -0.07 [-0.88 to 0.74] | -0.54 [-1.51 to 0.43] | -0.33 [-0.74 to 0.08]
  Knee Extension - Left - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Knee Extension - Left - Week 73 | -0.60 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.00 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.25 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.28 [-0.76 to 0.19]
  Knee Extension - Right - Baseline: number analyzed (Participants) | 16 | 17 | 18 | 51
  Knee Extension - Right - Baseline | 4.33 [3.09 to 5.58] | 4.48 [3.53 to 5.44] | 4.81 [3.16 to 6.46] | 4.55 [3.83 to 5.27]
  Knee Extension - Right - Week 13: number analyzed (Participants) | 16 | 17 | 17 | 50
  Knee Extension - Right - Week 13 | -0.35 [-1.26 to 0.56] | -0.13 [-0.89 to 0.63] | -0.93 [-1.82 to -0.03] | -0.47 [-0.94 to 0.00]
  Knee Extension - Right - Week 25: number analyzed (Participants) | 11 | 12 | 14 | 37
  Knee Extension - Right - Week 25 | -0.35 [-1.10 to 0.39] | -1.08 [-1.80 to -0.36] | -0.94 [-1.71 to -0.16] | -0.81 [-1.22 to -0.41]
  Knee Extension - Right - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Knee Extension - Right - Week 49 | -0.74 [-1.71 to 0.22] | -0.23 [-1.64 to 1.18] | -0.69 [-2.33 to 0.96] | -0.57 [-1.21 to 0.07]
  Knee Extension - Right - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Knee Extension - Right - Week 73 | -0.45 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.35 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.45 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.75 [-1.72 to 0.22]
  Shoulder Abduction - Left - Baseline: number analyzed (Participants) | 16 | 17 | 18 | 51
  Shoulder Abduction - Left - Baseline | 3.83 [2.83 to 4.83] | 3.95 [3.37 to 4.52] | 3.75 [3.08 to 4.42] | 3.84 [3.44 to 4.25]
  Shoulder Abduction - Left - Week 13: number analyzed (Participants) | 16 | 17 | 17 | 50
  Shoulder Abduction - Left - Week 13 | -0.14 [-0.71 to 0.43] | -0.31 [-0.95 to 0.34] | -0.28 [-0.69 to 0.14] | -0.24 [-0.54 to 0.05]
  Shoulder Abduction - Left - Week 25: number analyzed (Participants) | 11 | 12 | 14 | 37
  Shoulder Abduction - Left - Week 25 | -0.29 [-1.22 to 0.64] | -0.53 [-1.21 to 0.16] | -0.44 [-0.81 to -0.06] | -0.42 [-0.76 to -0.08]
  Shoulder Abduction - Left - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Shoulder Abduction - Left - Week 49 | -0.44 [-2.36 to 1.47] | -0.45 [-1.88 to 0.98] | -0.50 [-0.77 to -0.23] | -0.47 [-1.10 to 0.17]
  Shoulder Abduction - Left - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Shoulder Abduction - Left - Week 73 | -0.75 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.30 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.20 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.62 [-1.84 to 0.61]
  Shoulder Abduction - Right - Baseline: number analyzed (Participants) | 16 | 17 | 18 | 51
  Shoulder Abduction - Right - Baseline | 3.99 [2.72 to 5.26] | 4.26 [3.29 to 5.23] | 3.91 [3.10 to 4.71] | 4.05 [3.51 to 4.60]
  Shoulder Abduction - Right - Week 13: number analyzed (Participants) | 16 | 17 | 17 | 50
  Shoulder Abduction - Right - Week 13 | -0.16 [-0.75 to 0.44] | -0.55 [-1.50 to 0.40] | -0.39 [-0.96 to 0.18] | -0.37 [-0.76 to 0.02]
  Shoulder Abduction - Right - Week 25: number analyzed (Participants) | 11 | 12 | 14 | 37
  Shoulder Abduction - Right - Week 25 | -0.05 [-1.02 to 0.91] | -0.81 [-1.89 to 0.27] | -0.59 [-1.34 to 0.16] | -0.50 [-0.99 to -0.01]
  Shoulder Abduction - Right - Week 49: number analyzed (Participants) | 7 | 6 | 7 | 20
  Shoulder Abduction - Right - Week 49 | -0.49 [-2.95 to 1.98] | -0.60 [-1.78 to 0.58] | -0.16 [-0.58 to 0.27] | -0.41 [-1.17 to 0.36]
  Shoulder Abduction - Right - Week 73: number analyzed (Participants) | 2 | 2 | 2 | 6
  Shoulder Abduction - Right - Week 73 | -0.30 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.55 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.60 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.82 [-1.51 to -0.12]

48. Secondary Outcome: Change From Baseline on the Myometry Based Muscle Strength - Overall Baseline
Description: Muscle strength was quantified by means of a handheld dynamometer. The following muscle groups were evaluated: knee extension, elbow flexion, elbow extension, hip abduction and shoulder abduction. 95% Confidence Interval was not calculated when less than or equal to 3 participants' data were available.
  Overall baseline was defined as the last pre-dose assessment prior to the first day of dosing in study B5161002. Week 1 was start of the study treatment in parent study B5161002.
Time Frame: Baseline,Weeks 9,17,25,33,41,49,57,65,73,81,89,97,110,122,146,170.
Population: as for outcome 30
Measure: Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Kilograms
  Elbow Extension-Left - Baseline | 3.76 [2.48 to 5.05] | 3.51 [2.46 to 4.55] | 2.90 [2.25 to 3.55] | 3.38 [2.82 to 3.94]
  Elbow Extension-Left - Week 9: number analyzed (Participants) | 18 | 19 | 20 | 57
  Elbow Extension-Left - Week 9 | -0.10 [-0.67 to 0.47] | 0.76 [-0.09 to 1.61] | 0.20 [-0.09 to 0.48] | 0.29 [-0.05 to 0.63]
  Elbow Extension-Left - Week 17: number analyzed (Participants) | 19 | 19 | 20 | 58
  Elbow Extension-Left - Week 17 | 0.08 [-0.60 to 0.77] | -0.15 [-1.04 to 0.74] | 0.17 [-0.17 to 0.50] | 0.04 [-0.33 to 0.40]
  Elbow Extension-Left - Week 25: number analyzed (Participants) | 18 | 20 | 20 | 58
  Elbow Extension-Left - Week 25 | -0.74 [-1.75 to 0.26] | -0.03 [-1.07 to 1.01] | -0.02 [-0.30 to 0.26] | -0.25 [-0.71 to 0.21]
  Elbow Extension-Left - Week 33: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Extension-Left - Week 33 | -0.65 [-1.56 to 0.26] | -0.37 [-1.08 to 0.34] | 0.19 [-0.23 to 0.62] | -0.28 [-0.67 to 0.12]
  Elbow Extension-Left - Week 41: number analyzed (Participants) | 18 | 20 | 18 | 56
  Elbow Extension-Left - Week 41 | -0.43 [-1.82 to 0.96] | -0.20 [-1.04 to 0.64] | -0.02 [-0.36 to 0.33] | -0.22 [-0.73 to 0.30]
  Elbow Extension-Left - Week 49: number analyzed (Participants) | 19 | 19 | 19 | 57
  Elbow Extension-Left - Week 49 | -0.65 [-1.76 to 0.45] | -0.46 [-1.30 to 0.37] | 0.25 [-0.14 to 0.65] | -0.29 [-0.75 to 0.17]
  Elbow Extension-Left - Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Elbow Extension-Left - Week 57 | -0.75 [-1.77 to 0.26] | -0.60 [-1.41 to 0.21] | -0.01 [-0.31 to 0.30] | -0.46 [-0.90 to -0.03]
  Elbow Extension-Left - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Extension-Left - Week 65 | -0.70 [-1.62 to 0.22] | -0.30 [-1.36 to 0.76] | 0.12 [-0.25 to 0.48] | -0.29 [-0.76 to 0.17]
  Elbow Extension-Left - Week 73: number analyzed (Participants) | 18 | 20 | 20 | 58
  Elbow Extension-Left - Week 73 | -0.87 [-1.85 to 0.10] | -0.19 [-1.11 to 0.73] | 0.27 [-0.16 to 0.70] | -0.24 [-0.69 to 0.21]
  Elbow Extension-Left - Week 81: number analyzed (Participants) | 18 | 19 | 20 | 57
  Elbow Extension-Left - Week 81 | -0.75 [-1.65 to 0.15] | -0.44 [-1.21 to 0.33] | 0.22 [-0.17 to 0.61] | -0.31 [-0.70 to 0.09]
  Elbow Extension-Left - Week 89: number analyzed (Participants) | 16 | 20 | 19 | 55
  Elbow Extension-Left - Week 89 | -0.63 [-1.54 to 0.29] | -0.69 [-1.39 to 0.02] | 0.09 [-0.36 to 0.54] | -0.40 [-0.79 to -0.01]
  Elbow Extension-Left - Week 97 | -0.69 [-1.66 to 0.28] | -0.49 [-1.22 to 0.24] | -0.05 [-0.47 to 0.38] | -0.40 [-0.81 to 0.00]
  Elbow Extension-Left - Week 110: number analyzed (Participants) | 16 | 17 | 17 | 50
  Elbow Extension-Left - Week 110 | -0.99 [-2.00 to 0.01] | -1.08 [-2.21 to 0.05] | -0.36 [-0.84 to 0.12] | -0.81 [-1.31 to -0.31]
  Elbow Extension-Left - Week 122: number analyzed (Participants) | 11 | 12 | 14 | 37
  Elbow Extension-Left - Week 122 | -1.81 [-3.30 to -0.32] | -0.58 [-1.56 to 0.40] | 0.06 [-0.26 to 0.38] | -0.71 [-1.26 to -0.15]
  Elbow Extension-Left - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Elbow Extension-Left - Week 146 | -1.90 [-4.56 to 0.76] | -0.72 [-2.15 to 0.72] | 0.06 [-0.43 to 0.54] | -0.86 [-1.79 to 0.07]
  Elbow Extension-Left - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Elbow Extension-Left - Week 170 | -4.55 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.20 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.20 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.65 [-4.05 to 0.75]
  Elbow Extension-Right - Baseline | 3.85 [2.63 to 5.06] | 3.49 [2.31 to 4.67] | 2.96 [2.25 to 3.66] | 3.42 [2.85 to 4.00]
  Elbow Extension-Right - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Elbow Extension-Right - Week 9 | -0.43 [-1.11 to 0.25] | 0.77 [-0.28 to 1.82] | 0.26 [-0.02 to 0.53] | 0.20 [-0.22 to 0.62]
  Elbow Extension-Right - Week 17: number analyzed (Participants) | 19 | 19 | 20 | 58
  Elbow Extension-Right - Week 17 | 0.03 [-0.88 to 0.93] | 0.08 [-1.02 to 1.19] | 0.30 [0.00 to 0.59] | 0.14 [-0.31 to 0.59]
  Elbow Extension-Right - Week 25 | -0.64 [-1.54 to 0.27] | 0.13 [-0.91 to 1.16] | 0.27 [0.03 to 0.51] | -0.07 [-0.52 to 0.38]
  Elbow Extension-Right - Week 33: number analyzed (Participants) | 18 | 20 | 19 | 57
  Elbow Extension-Right - Week 33 | -0.74 [-1.77 to 0.29] | -0.39 [-1.22 to 0.45] | 0.20 [-0.18 to 0.58] | -0.30 [-0.74 to 0.14]
  Elbow Extension-Right - Week 41: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Extension-Right - Week 41 | -0.61 [-1.74 to 0.52] | -0.44 [-1.22 to 0.35] | -0.12 [-0.47 to 0.24] | -0.39 [-0.84 to 0.06]
  Elbow Extension-Right - Week 49: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Extension-Right - Week 49 | -0.56 [-1.68 to 0.56] | -0.45 [-1.27 to 0.38] | 0.04 [-0.25 to 0.33] | -0.32 [-0.77 to 0.13]
  Elbow Extension-Right - Week 57: number analyzed (Participants) | 18 | 20 | 18 | 56
  Elbow Extension-Right - Week 57 | -1.01 [-1.98 to -0.04] | -0.65 [-1.50 to 0.21] | 0.09 [-0.18 to 0.36] | -0.53 [-0.96 to -0.09]
  Elbow Extension-Right - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Extension-Right - Week 65 | -0.88 [-1.85 to 0.09] | -0.20 [-1.34 to 0.94] | 0.28 [-0.14 to 0.71] | -0.26 [-0.77 to 0.24]
  Elbow Extension-Right - Week 73 | -1.07 [-2.08 to -0.07] | -0.26 [-1.36 to 0.85] | 0.17 [-0.23 to 0.57] | -0.37 [-0.88 to 0.13]
  Elbow Extension-Right - Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Elbow Extension-Right - Week 81 | -0.71 [-1.68 to 0.27] | -0.67 [-1.61 to 0.26] | 0.59 [0.18 to 0.99] | -0.25 [-0.71 to 0.21]
  Elbow Extension-Right - Week 89: number analyzed (Participants) | 17 | 20 | 19 | 56
  Elbow Extension-Right - Week 89 | -1.00 [-2.08 to 0.08] | -0.58 [-1.40 to 0.24] | 0.17 [-0.23 to 0.57] | -0.45 [-0.90 to -0.01]
  Elbow Extension-Right - Week 97 | -0.76 [-1.76 to 0.24] | -0.48 [-1.50 to 0.54] | -0.04 [-0.38 to 0.31] | -0.42 [-0.88 to 0.04]
  Elbow Extension-Right - Week 110: number analyzed (Participants) | 16 | 17 | 17 | 50
  Elbow Extension-Right - Week 110 | -1.12 [-2.21 to -0.03] | -0.94 [-2.10 to 0.23] | -0.38 [-0.92 to 0.17] | -0.80 [-1.33 to -0.28]
  Elbow Extension-Right - Week 122: number analyzed (Participants) | 10 | 12 | 14 | 36
  Elbow Extension-Right - Week 122 | -1.77 [-3.53 to -0.01] | -0.63 [-1.25 to -0.02] | 0.14 [-0.34 to 0.61] | -0.65 [-1.21 to -0.09]
  Elbow Extension-Right - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Elbow Extension-Right - Week 146 | -1.70 [-4.42 to 1.02] | -0.75 [-1.06 to -0.44] | -0.03 [-0.74 to 0.68] | -0.83 [-1.70 to 0.04]
  Elbow Extension-Right - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Elbow Extension-Right - Week 170 | -4.35 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.45 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.15 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.98 [-4.01 to 0.04]
  Elbow Flexion-Left - Baseline | 4.58 [2.96 to 6.19] | 4.21 [3.14 to 5.27] | 3.83 [3.01 to 4.64] | 4.20 [3.54 to 4.85]
  Elbow Flexion-Left - Week 9: number analyzed (Participants) | 18 | 19 | 20 | 57
  Elbow Flexion-Left - Week 9 | -0.11 [-1.17 to 0.95] | 1.06 [-0.01 to 2.14] | 0.01 [-0.46 to 0.47] | 0.32 [-0.18 to 0.82]
  Elbow Flexion-Left -Week 17: number analyzed (Participants) | 19 | 19 | 20 | 58
  Elbow Flexion-Left -Week 17 | -0.37 [-1.69 to 0.95] | -0.05 [-0.82 to 0.72] | -0.05 [-0.56 to 0.47] | -0.15 [-0.65 to 0.35]
  Elbow Flexion-Left - Week 25: number analyzed (Participants) | 18 | 20 | 20 | 58
  Elbow Flexion-Left - Week 25 | -0.72 [-2.29 to 0.85] | 0.02 [-1.05 to 1.09] | -0.06 [-0.48 to 0.37] | -0.24 [-0.83 to 0.36]
  Elbow Flexion-Left - Week 33: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Flexion-Left - Week 33 | -0.59 [-1.97 to 0.79] | -0.45 [-1.10 to 0.20] | -0.04 [-0.41 to 0.34] | -0.36 [-0.85 to 0.13]
  Elbow Flexion-Left - Week 41: number analyzed (Participants) | 18 | 20 | 18 | 56
  Elbow Flexion-Left - Week 41 | -0.77 [-2.40 to 0.87] | -0.41 [-1.11 to 0.29] | -0.34 [-0.75 to 0.06] | -0.50 [-1.06 to 0.06]
  Elbow Flexion-Left - Week 49: number analyzed (Participants) | 19 | 19 | 19 | 57
  Elbow Flexion-Left - Week 49 | -1.12 [-2.41 to 0.18] | -0.66 [-1.36 to 0.04] | -0.18 [-0.76 to 0.40] | -0.65 [-1.16 to -0.15]
  Elbow Flexion-Left - Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Elbow Flexion-Left - Week 57 | -1.02 [-2.43 to 0.39] | -0.57 [-1.27 to 0.14] | -0.29 [-0.75 to 0.16] | -0.63 [-1.15 to -0.11]
  Elbow Flexion-Left - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Flexion-Left - Week 65 | -1.01 [-2.39 to 0.38] | -0.67 [-1.52 to 0.18] | -0.20 [-0.60 to 0.20] | -0.63 [-1.15 to -0.10]
  Elbow Flexion-Left - Week 73: number analyzed (Participants) | 18 | 20 | 20 | 58
  Elbow Flexion-Left - Week 73 | -1.10 [-2.44 to 0.24] | -0.36 [-1.22 to 0.51] | -0.24 [-0.95 to 0.47] | -0.55 [-1.08 to -0.01]
  Elbow Flexion-Left - Week 81: number analyzed (Participants) | 18 | 19 | 20 | 57
  Elbow Flexion-Left - Week 81 | -0.91 [-2.28 to 0.46] | -0.62 [-1.37 to 0.13] | -0.19 [-0.65 to 0.28] | -0.56 [-1.06 to -0.06]
  Elbow Flexion-Left - Week 89: number analyzed (Participants) | 16 | 19 | 19 | 54
  Elbow Flexion-Left - Week 89 | -0.84 [-2.19 to 0.51] | -0.84 [-1.58 to -0.11] | -0.35 [-0.85 to 0.15] | -0.67 [-1.14 to -0.19]
  Elbow Flexion-Left - Week 97 | -0.71 [-2.24 to 0.82] | -0.68 [-1.56 to 0.20] | -0.55 [-1.20 to 0.11] | -0.64 [-1.22 to -0.06]
  Elbow Flexion-Left - Week 110: number analyzed (Participants) | 16 | 17 | 17 | 50
  Elbow Flexion-Left - Week 110 | -1.28 [-2.94 to 0.38] | -1.01 [-2.13 to 0.11] | -1.05 [-1.77 to -0.34] | -1.11 [-1.76 to -0.47]
  Elbow Flexion-Left - Week 122: number analyzed (Participants) | 11 | 12 | 14 | 37
  Elbow Flexion-Left - Week 122 | -2.32 [-4.57 to -0.06] | -0.95 [-2.06 to 0.16] | -0.61 [-1.13 to -0.08] | -1.23 [-1.97 to -0.49]
  Elbow Flexion-Left - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Elbow Flexion-Left - Week 146 | -1.94 [-4.63 to 0.75] | -0.42 [-2.43 to 1.60] | -0.53 [-1.46 to 0.41] | -0.99 [-1.98 to 0.00]
  Elbow Flexion-Left - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Elbow Flexion-Left - Week 170 | -4.70 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.25 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.25 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -2.40 [-4.30 to -0.50]
  Elbow Flexion-Right - Baseline | 4.66 [3.43 to 5.89] | 4.24 [3.18 to 5.30] | 3.73 [2.93 to 4.53] | 4.20 [3.63 to 4.77]
  Elbow Flexion-Right - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Elbow Flexion-Right - Week 9 | -0.47 [-1.39 to 0.45] | 0.65 [-0.19 to 1.48] | 0.49 [-0.02 to 1.00] | 0.23 [-0.21 to 0.66]
  Elbow Flexion-Right - Week 17: number analyzed (Participants) | 19 | 19 | 20 | 58
  Elbow Flexion-Right - Week 17 | 0.09 [-0.83 to 1.02] | -0.08 [-0.97 to 0.80] | 0.11 [-0.23 to 0.45] | 0.04 [-0.37 to 0.45]
  Elbow Flexion-Right - Week 25 | -0.67 [-1.58 to 0.24] | -0.14 [-1.20 to 0.92] | 0.00 [-0.44 to 0.44] | -0.26 [-0.73 to 0.20]
  Elbow Flexion-Right - Week 33: number analyzed (Participants) | 18 | 20 | 19 | 57
  Elbow Flexion-Right - Week 33 | -0.56 [-1.57 to 0.46] | -0.36 [-1.00 to 0.29] | 0.06 [-0.40 to 0.52] | -0.28 [-0.68 to 0.12]
  Elbow Flexion-Right - Week 41: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Flexion-Right - Week 41 | -0.60 [-1.90 to 0.70] | -0.29 [-0.95 to 0.38] | -0.26 [-0.70 to 0.18] | -0.38 [-0.85 to 0.09]
  Elbow Flexion-Right - Week 49: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Flexion-Right - Week 49 | -0.73 [-1.74 to 0.28] | -0.66 [-1.24 to -0.07] | -0.01 [-0.48 to 0.47] | -0.47 [-0.87 to -0.07]
  Elbow Flexion-Right - Week 57: number analyzed (Participants) | 18 | 20 | 18 | 56
  Elbow Flexion-Right - Week 57 | -1.11 [-2.15 to -0.07] | -0.42 [-0.97 to 0.13] | -0.23 [-0.65 to 0.19] | -0.58 [-0.98 to -0.18]
  Elbow Flexion-Right - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Elbow Flexion-Right - Week 65 | -0.77 [-1.72 to 0.18] | -0.33 [-1.09 to 0.43] | -0.06 [-0.50 to 0.37] | -0.39 [-0.80 to 0.02]
  Elbow Flexion-Right - Week 73 | -0.93 [-1.80 to -0.06] | -0.31 [-1.03 to 0.41] | -0.11 [-0.68 to 0.46] | -0.44 [-0.85 to -0.04]
  Elbow Flexion-Right - Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Elbow Flexion-Right - Week 81 | -0.99 [-1.87 to -0.12] | -0.30 [-0.96 to 0.36] | 0.03 [-0.48 to 0.53] | -0.42 [-0.81 to -0.02]
  Elbow Flexion-Right - Week 89: number analyzed (Participants) | 18 | 19 | 19 | 56
  Elbow Flexion-Right - Week 89 | -0.87 [-1.77 to 0.04] | -0.58 [-1.18 to 0.02] | -0.17 [-0.59 to 0.25] | -0.53 [-0.90 to -0.17]
  Elbow Flexion-Right - Week 97 | -0.86 [-1.93 to 0.20] | -0.35 [-1.13 to 0.44] | -0.57 [-1.19 to 0.06] | -0.59 [-1.04 to -0.13]
  Elbow Flexion-Right - Week 110: number analyzed (Participants) | 16 | 17 | 17 | 50
  Elbow Flexion-Right - Week 110 | -1.30 [-2.44 to -0.16] | -1.22 [-2.29 to -0.16] | -0.85 [-1.46 to -0.25] | -1.12 [-1.64 to -0.61]
  Elbow Flexion-Right - Week 122: number analyzed (Participants) | 10 | 12 | 14 | 36
  Elbow Flexion-Right - Week 122 | -2.34 [-4.28 to -0.40] | -0.91 [-2.08 to 0.27] | -0.06 [-0.65 to 0.52] | -0.98 [-1.67 to -0.28]
  Elbow Flexion-Right - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Elbow Flexion-Right - Week 146 | -2.00 [-4.72 to 0.72] | -0.90 [-2.00 to 0.20] | -0.63 [-1.26 to 0.00] | -1.19 [-2.07 to -0.31]
  Elbow Flexion-Right - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Elbow Flexion-Right - Week 170 | -5.35 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.20 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.15 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -2.57 [-4.87 to -0.26]
  Hip Abduction-Left - Baseline | 4.31 [3.23 to 5.38] | 5.10 [3.84 to 6.36] | 4.35 [3.56 to 5.13] | 4.59 [4.01 to 5.17]
  Hip Abduction-Left - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Hip Abduction-Left - Week 9 | 0.23 [-0.86 to 1.32] | 1.19 [0.17 to 2.21] | 0.38 [-0.25 to 1.01] | 0.60 [0.08 to 1.11]
  Hip Abduction-Left - Week 17: number analyzed (Participants) | 19 | 19 | 20 | 58
  Hip Abduction-Left - Week 17 | 0.36 [-0.94 to 1.65] | -0.03 [-1.10 to 1.04] | 0.74 [0.10 to 1.37] | 0.36 [-0.20 to 0.92]
  Hip Abduction-Left - Week 25: number analyzed (Participants) | 19 | 20 | 19 | 58
  Hip Abduction-Left - Week 25 | -0.49 [-1.85 to 0.87] | 0.41 [-0.76 to 1.58] | 0.52 [-0.13 to 1.16] | 0.15 [-0.46 to 0.76]
  Hip Abduction-Left - Week 33: number analyzed (Participants) | 19 | 20 | 19 | 58
  Hip Abduction-Left - Week 33 | 0.18 [-1.16 to 1.51] | 0.13 [-0.85 to 1.11] | 0.26 [-0.47 to 0.99] | 0.19 [-0.38 to 0.75]
  Hip Abduction-Left - Week 41: number analyzed (Participants) | 17 | 20 | 19 | 56
  Hip Abduction-Left - Week 41 | -0.64 [-1.66 to 0.37] | -0.19 [-1.14 to 0.77] | 0.59 [-0.08 to 1.27] | -0.06 [-0.56 to 0.44]
  Hip Abduction-Left - Week 49: number analyzed (Participants) | 19 | 20 | 19 | 58
  Hip Abduction-Left - Week 49 | 0.56 [-1.16 to 2.27] | -0.47 [-1.27 to 0.34] | 0.55 [-0.29 to 1.38] | 0.20 [-0.45 to 0.85]
  Hip Abduction-Left - Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Hip Abduction-Left - Week 57 | -0.16 [-1.11 to 0.79] | -0.06 [-0.89 to 0.77] | 0.62 [-0.06 to 1.29] | 0.12 [-0.34 to 0.58]
  Hip Abduction-Left - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Hip Abduction-Left - Week 65 | -0.24 [-1.19 to 0.71] | -0.06 [-1.10 to 0.98] | 0.86 [0.03 to 1.68] | 0.18 [-0.35 to 0.71]
  Hip Abduction-Left - Week 73: number analyzed (Participants) | 18 | 20 | 20 | 58
  Hip Abduction-Left - Week 73 | 0.00 [-1.04 to 1.04] | 0.31 [-0.81 to 1.43] | 1.06 [0.07 to 2.04] | 0.47 [-0.11 to 1.05]
  Hip Abduction-Left - Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Hip Abduction-Left - Week 81 | -0.43 [-1.32 to 0.46] | 0.17 [-0.91 to 1.26] | 1.35 [0.63 to 2.06] | 0.38 [-0.15 to 0.91]
  Hip Abduction-Left - Week 89: number analyzed (Participants) | 18 | 20 | 19 | 57
  Hip Abduction-Left - Week 89 | 0.37 [-0.64 to 1.38] | 0.14 [-0.86 to 1.13] | 0.78 [-0.01 to 1.57] | 0.42 [-0.09 to 0.94]
  Hip Abduction-Left - Week 97 | -0.11 [-1.02 to 0.81] | -0.07 [-1.28 to 1.14] | 0.40 [-0.25 to 1.05] | 0.08 [-0.44 to 0.60]
  Hip Abduction-Left - Week 110: number analyzed (Participants) | 16 | 17 | 16 | 49
  Hip Abduction-Left - Week 110 | -0.18 [-1.41 to 1.04] | -0.68 [-2.16 to 0.79] | 0.22 [-0.92 to 1.36] | -0.22 [-0.93 to 0.48]
  Hip Abduction-Left - Week 122: number analyzed (Participants) | 10 | 12 | 13 | 35
  Hip Abduction-Left - Week 122 | -0.09 [-2.41 to 2.23] | -0.13 [-1.61 to 1.36] | 0.58 [-0.29 to 1.46] | 0.15 [-0.65 to 0.95]
  Hip Abduction-Left - Week 146: number analyzed (Participants) | 7 | 5 | 7 | 19
  Hip Abduction-Left - Week 146 | -1.24 [-4.04 to 1.55] | -0.26 [-2.36 to 1.84] | 0.84 [-0.84 to 2.53] | -0.22 [-1.36 to 0.93]
  Hip Abduction-Left - Week 170: number analyzed (Participants) | 2 | 2 | 1 | 5
  Hip Abduction-Left - Week 170 | -4.75 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -2.00 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.50 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -2.80 [-5.16 to -0.44]
  Hip Abduction-Right - Baseline | 4.14 [3.05 to 5.22] | 5.39 [3.95 to 6.83] | 4.53 [3.30 to 5.75] | 4.69 [3.99 to 5.39]
  Hip Abduction-Right - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Hip Abduction-Right - Week 9 | 0.56 [-0.84 to 1.97] | 1.05 [-0.03 to 2.13] | 0.03 [-0.61 to 0.67] | 0.54 [-0.05 to 1.13]
  Hip Abduction-Right - Week 17: number analyzed (Participants) | 19 | 19 | 20 | 58
  Hip Abduction-Right - Week 17 | 0.56 [-0.62 to 1.75] | -0.51 [-1.67 to 0.66] | 0.46 [-0.22 to 1.13] | 0.18 [-0.39 to 0.74]
  Hip Abduction-Right - Week 25 | -0.31 [-1.44 to 0.83] | -0.23 [-1.57 to 1.11] | 0.47 [-0.11 to 1.05] | -0.02 [-0.60 to 0.57]
  Hip Abduction-Right - Week 33: number analyzed (Participants) | 19 | 20 | 19 | 58
  Hip Abduction-Right - Week 33 | 0.42 [-1.09 to 1.93] | -0.80 [-1.89 to 0.29] | 0.12 [-0.80 to 1.04] | -0.10 [-0.76 to 0.56]
  Hip Abduction-Right - Week 41: number analyzed (Participants) | 18 | 20 | 19 | 57
  Hip Abduction-Right - Week 41 | -0.18 [-1.46 to 1.10] | -0.60 [-1.48 to 0.28] | 0.22 [-0.60 to 1.03] | -0.19 [-0.74 to 0.35]
  Hip Abduction-Right - Week 49: number analyzed (Participants) | 19 | 20 | 19 | 58
  Hip Abduction-Right - Week 49 | 0.92 [-0.74 to 2.58] | -0.67 [-1.71 to 0.38] | 0.33 [-0.38 to 1.03] | 0.18 [-0.49 to 0.85]
  Hip Abduction-Right - Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Hip Abduction-Right - Week 57 | 0.13 [-0.91 to 1.16] | -0.63 [-1.66 to 0.41] | 0.08 [-0.65 to 0.80] | -0.15 [-0.68 to 0.37]
  Hip Abduction-Right - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Hip Abduction-Right - Week 65 | 0.19 [-0.82 to 1.20] | -0.17 [-1.52 to 1.18] | 0.75 [0.10 to 1.40] | 0.25 [-0.33 to 0.83]
  Hip Abduction-Right - Week 73 | 0.12 [-0.87 to 1.10] | 0.04 [-1.34 to 1.41] | 0.73 [0.03 to 1.42] | 0.29 [-0.28 to 0.87]
  Hip Abduction-Right - Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Hip Abduction-Right - Week 81 | 0.03 [-0.97 to 1.02] | -0.62 [-1.62 to 0.38] | 0.69 [-0.01 to 1.38] | 0.04 [-0.47 to 0.55]
  Hip Abduction-Right - Week 89: number analyzed (Participants) | 18 | 20 | 19 | 57
  Hip Abduction-Right - Week 89 | 0.08 [-0.72 to 0.87] | -0.44 [-1.41 to 0.54] | 0.68 [0.08 to 1.28] | 0.10 [-0.36 to 0.56]
  Hip Abduction-Right - Week 97 | 0.05 [-0.96 to 1.06] | -0.20 [-1.43 to 1.03] | 0.18 [-0.93 to 1.29] | 0.01 [-0.60 to 0.62]
  Hip Abduction-Right - Week 110: number analyzed (Participants) | 16 | 17 | 16 | 49
  Hip Abduction-Right - Week 110 | 0.04 [-0.96 to 1.05] | -1.06 [-2.77 to 0.66] | -0.23 [-1.79 to 1.33] | -0.43 [-1.23 to 0.37]
  Hip Abduction-Right - Week 122: number analyzed (Participants) | 10 | 12 | 13 | 35
  Hip Abduction-Right - Week 122 | -0.07 [-2.54 to 2.40] | -0.77 [-2.37 to 0.84] | 0.52 [-0.52 to 1.56] | -0.09 [-0.97 to 0.79]
  Hip Abduction-Right - Week 146: number analyzed (Participants) | 7 | 5 | 7 | 19
  Hip Abduction-Right - Week 146 | -1.10 [-3.32 to 1.12] | -1.44 [-2.89 to 0.01] | 1.13 [0.25 to 2.01] | -0.37 [-1.32 to 0.59]
  Hip Abduction-Right - Week 170: number analyzed (Participants) | 2 | 2 | 1 | 5
  Hip Abduction-Right - Week 170 | -4.30 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.75 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 1.60 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -2.10 [-5.12 to 0.92]
  Knee Extension-Left - Baseline | 5.99 [4.01 to 7.98] | 5.38 [4.01 to 6.74] | 5.21 [3.53 to 6.88] | 5.52 [4.60 to 6.43]
  Knee Extension-Left - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Knee Extension-Left - Week 9 | -0.54 [-1.56 to 0.48] | 1.20 [-0.24 to 2.64] | -0.16 [-0.81 to 0.49] | 0.16 [-0.45 to 0.77]
  Knee Extension-Left - Week 17: number analyzed (Participants) | 19 | 19 | 20 | 58
  Knee Extension-Left - Week 17 | -0.88 [-2.29 to 0.53] | 0.17 [-0.95 to 1.29] | -0.12 [-0.77 to 0.54] | -0.27 [-0.88 to 0.33]
  Knee Extension-Left - Week 25: number analyzed (Participants) | 19 | 20 | 19 | 58
  Knee Extension-Left - Week 25 | -1.66 [-2.98 to -0.34] | -0.14 [-1.37 to 1.09] | -0.38 [-0.84 to 0.07] | -0.72 [-1.33 to -0.11]
  Knee Extension-Left - Week 33: number analyzed (Participants) | 19 | 20 | 19 | 58
  Knee Extension-Left - Week 33 | -1.35 [-3.13 to 0.43] | -0.54 [-1.41 to 0.33] | -0.55 [-1.19 to 0.10] | -0.81 [-1.46 to -0.16]
  Knee Extension-Left - Week 41: number analyzed (Participants) | 17 | 20 | 19 | 56
  Knee Extension-Left - Week 41 | -1.53 [-3.47 to 0.41] | -0.87 [-1.84 to 0.11] | -0.67 [-1.14 to -0.21] | -1.00 [-1.66 to -0.34]
  Knee Extension-Left - Week 49: number analyzed (Participants) | 19 | 20 | 19 | 58
  Knee Extension-Left - Week 49 | -1.27 [-3.24 to 0.71] | -0.59 [-1.48 to 0.30] | -0.85 [-1.50 to -0.20] | -0.90 [-1.60 to -0.19]
  Knee Extension-Left - Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Knee Extension-Left - Week 57 | -1.67 [-3.50 to 0.16] | -0.77 [-1.80 to 0.27] | -0.73 [-1.79 to 0.32] | -1.06 [-1.80 to -0.31]
  Knee Extension-Left - Week 65: number analyzed (Participants) | 18 | 20 | 19 | 57
  Knee Extension-Left - Week 65 | -1.23 [-2.88 to 0.41] | -0.46 [-1.68 to 0.76] | -0.42 [-1.31 to 0.47] | -0.69 [-1.39 to 0.01]
  Knee Extension-Left - Week 73: number analyzed (Participants) | 18 | 20 | 20 | 58
  Knee Extension-Left - Week 73 | -1.78 [-3.77 to 0.21] | -0.39 [-1.85 to 1.07] | -0.02 [-0.57 to 0.53] | -0.69 [-1.48 to 0.10]
  Knee Extension-Left - Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Knee Extension-Left - Week 81 | -1.99 [-3.74 to -0.25] | -1.52 [-2.51 to -0.53] | -0.23 [-1.03 to 0.58] | -1.23 [-1.93 to -0.53]
  Knee Extension-Left - Week 89: number analyzed (Participants) | 18 | 20 | 19 | 57
  Knee Extension-Left - Week 89 | -2.16 [-3.98 to -0.33] | -1.45 [-2.46 to -0.43] | -0.27 [-1.16 to 0.61] | -1.28 [-2.00 to -0.56]
  Knee Extension-Left - Week 97 | -1.80 [-3.65 to 0.05] | -1.24 [-2.41 to -0.07] | -0.82 [-1.93 to 0.30] | -1.28 [-2.04 to -0.51]
  Knee Extension-Left - Week 110: number analyzed (Participants) | 16 | 17 | 17 | 50
  Knee Extension-Left - Week 110 | -2.28 [-4.26 to -0.30] | -1.79 [-3.16 to -0.42] | -1.89 [-3.18 to -0.60] | -1.98 [-2.82 to -1.15]
  Knee Extension-Left - Week 122: number analyzed (Participants) | 11 | 12 | 14 | 37
  Knee Extension-Left - Week 122 | -3.31 [-6.35 to -0.27] | -2.03 [-3.46 to -0.59] | -1.04 [-1.63 to -0.46] | -2.04 [-3.01 to -1.06]
  Knee Extension-Left - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Knee Extension-Left - Week 146 | -3.36 [-8.02 to 1.31] | -0.83 [-1.93 to 0.26] | -0.57 [-1.50 to 0.36] | -1.63 [-3.13 to -0.12]
  Knee Extension-Left - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Knee Extension-Left - Week 170 | -7.10 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.45 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.30 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -2.62 [-6.43 to 1.20]
  Knee Extension-Right - Baseline | 6.12 [4.21 to 8.04] | 5.91 [4.43 to 7.39] | 5.08 [3.31 to 6.85] | 5.70 [4.76 to 6.64]
  Knee Extension-Right - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Knee Extension-Right - Week 9 | -0.24 [-1.37 to 0.88] | 1.02 [-0.49 to 2.53] | 0.08 [-0.51 to 0.66] | 0.28 [-0.34 to 0.90]
  Knee Extension-Right - Week 17: number analyzed (Participants) | 19 | 19 | 20 | 58
  Knee Extension-Right - Week 17 | -0.70 [-1.86 to 0.46] | -0.26 [-1.33 to 0.81] | -0.16 [-0.85 to 0.53] | -0.37 [-0.91 to 0.17]
  Knee Extension-Right - Week 25 | -1.27 [-2.92 to 0.37] | -0.71 [-2.06 to 0.64] | -0.21 [-0.82 to 0.40] | -0.72 [-1.42 to -0.03]
  Knee Extension-Right - Week 33: number analyzed (Participants) | 19 | 20 | 19 | 58
  Knee Extension-Right - Week 33 | -0.74 [-2.63 to 1.15] | -0.91 [-1.94 to 0.12] | -0.39 [-1.08 to 0.31] | -0.68 [-1.39 to 0.02]
  Knee Extension-Right - Week 41: number analyzed (Participants) | 17 | 20 | 19 | 56
  Knee Extension-Right - Week 41 | -1.16 [-3.13 to 0.80] | -1.07 [-2.19 to 0.05] | -0.28 [-0.96 to 0.40] | -0.83 [-1.54 to -0.12]
  Knee Extension-Right - Week 49: number analyzed (Participants) | 19 | 20 | 19 | 58
  Knee Extension-Right - Week 49 | -1.23 [-3.10 to 0.65] | -1.04 [-2.00 to -0.08] | -0.34 [-0.90 to 0.22] | -0.87 [-1.55 to -0.19]
  Knee Extension-Right - Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Knee Extension-Right - Week 57 | -1.44 [-3.16 to 0.28] | -1.16 [-2.24 to -0.08] | -0.69 [-1.45 to 0.06] | -1.11 [-1.79 to -0.42]
  Knee Extension-Right - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Knee Extension-Right - Week 65 | -1.28 [-2.84 to 0.28] | -1.12 [-2.44 to 0.20] | -0.26 [-1.39 to 0.87] | -0.89 [-1.63 to -0.15]
  Knee Extension-Right - Week 73 | -1.57 [-3.28 to 0.14] | -1.24 [-2.55 to 0.08] | 0.15 [-0.41 to 0.70] | -0.87 [-1.59 to -0.16]
  Knee Extension-Right - Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Knee Extension-Right - Week 81 | -1.82 [-3.37 to -0.26] | -1.97 [-3.11 to -0.84] | 0.08 [-0.67 to 0.82] | -1.22 [-1.90 to -0.53]
  Knee Extension-Right - Week 89: number analyzed (Participants) | 18 | 20 | 19 | 57
  Knee Extension-Right - Week 89 | -2.05 [-3.88 to -0.22] | -1.80 [-2.83 to -0.76] | -0.21 [-0.87 to 0.45] | -1.35 [-2.05 to -0.64]
  Knee Extension-Right - Week 97 | -1.73 [-3.43 to -0.02] | -1.79 [-2.95 to -0.62] | -0.44 [-1.87 to 1.00] | -1.31 [-2.11 to -0.51]
  Knee Extension-Right - Week 110: number analyzed (Participants) | 16 | 17 | 17 | 50
  Knee Extension-Right - Week 110 | -2.21 [-3.84 to -0.58] | -2.05 [-3.48 to -0.63] | -1.42 [-2.72 to -0.12] | -1.89 [-2.67 to -1.11]
  Knee Extension-Right - Week 122: number analyzed (Participants) | 11 | 12 | 14 | 37
  Knee Extension-Right - Week 122 | -2.77 [-5.29 to -0.26] | -2.78 [-4.36 to -1.19] | -0.44 [-1.19 to 0.31] | -1.89 [-2.82 to -0.97]
  Knee Extension-Right - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Knee Extension-Right - Week 146 | -3.21 [-7.01 to 0.58] | -1.13 [-2.61 to 0.34] | -0.56 [-1.86 to 0.75] | -1.66 [-2.97 to -0.35]
  Knee Extension-Right - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Knee Extension-Right - Week 170 | -7.35 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -2.00 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.75 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -3.37 [-6.71 to -0.02]
  Shoulder Abduction-Left - Baseline | 3.55 [2.66 to 4.45] | 4.24 [3.26 to 5.22] | 3.44 [2.71 to 4.17] | 3.75 [3.26 to 4.23]
  Shoulder Abduction-Left - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Shoulder Abduction-Left - Week 9 | -0.01 [-0.78 to 0.76] | 0.58 [-0.21 to 1.38] | 0.08 [-0.44 to 0.59] | 0.21 [-0.17 to 0.60]
  Shoulder Abduction-Left - Week 17: number analyzed (Participants) | 19 | 19 | 20 | 58
  Shoulder Abduction-Left - Week 17 | 0.38 [-0.41 to 1.16] | -0.08 [-0.84 to 0.68] | 0.11 [-0.32 to 0.54] | 0.13 [-0.23 to 0.50]
  Shoulder Abduction-Left - Week 25 | -0.25 [-0.97 to 0.47] | 0.08 [-0.78 to 0.94] | 0.25 [-0.15 to 0.64] | 0.03 [-0.35 to 0.41]
  Shoulder Abduction-Left - Week 33: number analyzed (Participants) | 19 | 20 | 19 | 58
  Shoulder Abduction-Left - Week 33 | 0.09 [-1.01 to 1.19] | -0.20 [-0.95 to 0.56] | 0.12 [-0.11 to 0.35] | 0.00 [-0.42 to 0.42]
  Shoulder Abduction-Left - Week 41: number analyzed (Participants) | 18 | 20 | 18 | 56
  Shoulder Abduction-Left - Week 41 | 0.14 [-0.94 to 1.23] | -0.22 [-0.90 to 0.46] | 0.07 [-0.25 to 0.39] | -0.01 [-0.42 to 0.40]
  Shoulder Abduction-Left - Week 49: number analyzed (Participants) | 19 | 19 | 19 | 57
  Shoulder Abduction-Left - Week 49 | 0.36 [-0.97 to 1.69] | -0.29 [-0.90 to 0.31] | 0.19 [-0.19 to 0.58] | 0.09 [-0.39 to 0.56]
  Shoulder Abduction-Left - Week 57: number analyzed (Participants) | 19 | 20 | 18 | 57
  Shoulder Abduction-Left - Week 57 | -0.05 [-0.88 to 0.77] | -0.49 [-1.11 to 0.13] | 0.34 [-0.06 to 0.73] | -0.08 [-0.44 to 0.28]
  Shoulder Abduction-Left - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Shoulder Abduction-Left - Week 65 | -0.20 [-0.97 to 0.57] | 0.03 [-0.96 to 1.02] | 0.63 [0.26 to 0.99] | 0.15 [-0.27 to 0.57]
  Shoulder Abduction-Left - Week 73: number analyzed (Participants) | 18 | 20 | 20 | 58
  Shoulder Abduction-Left - Week 73 | -0.14 [-0.89 to 0.60] | 0.13 [-0.72 to 0.97] | 0.55 [0.19 to 0.90] | 0.19 [-0.19 to 0.56]
  Shoulder Abduction-Left - Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Shoulder Abduction-Left - Week 81 | -0.10 [-0.77 to 0.57] | -0.29 [-0.98 to 0.40] | 0.58 [0.27 to 0.89] | 0.07 [-0.25 to 0.40]
  Shoulder Abduction-Left - Week 89: number analyzed (Participants) | 17 | 20 | 19 | 56
  Shoulder Abduction-Left - Week 89 | 0.02 [-0.61 to 0.65] | -0.32 [-0.94 to 0.30] | 0.23 [-0.12 to 0.57] | -0.03 [-0.33 to 0.27]
  Shoulder Abduction-Left - Week 97 | 0.07 [-0.64 to 0.78] | -0.32 [-1.08 to 0.44] | 0.33 [-0.30 to 0.96] | 0.03 [-0.36 to 0.41]
  Shoulder Abduction-Left - Week 110: number analyzed (Participants) | 16 | 17 | 17 | 50
  Shoulder Abduction-Left - Week 110 | -0.06 [-0.99 to 0.87] | -0.86 [-2.02 to 0.30] | -0.01 [-0.55 to 0.53] | -0.32 [-0.82 to 0.19]
  Shoulder Abduction-Left - Week 122: number analyzed (Participants) | 11 | 12 | 14 | 37
  Shoulder Abduction-Left - Week 122 | -0.53 [-2.12 to 1.07] | -0.48 [-1.38 to 0.42] | 0.24 [-0.22 to 0.69] | -0.22 [-0.76 to 0.31]
  Shoulder Abduction-Left - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Shoulder Abduction-Left - Week 146 | -0.89 [-3.08 to 1.31] | -0.48 [-2.23 to 1.27] | -0.16 [-0.64 to 0.33] | -0.51 [-1.28 to 0.26]
  Shoulder Abduction-Left - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Shoulder Abduction-Left - Week 170 | -3.75 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.90 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | 0.85 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.27 [-3.62 to 1.09]
  Shoulder Abduction-Right - Baseline | 3.80 [2.81 to 4.79] | 4.33 [3.34 to 5.31] | 3.46 [2.76 to 4.16] | 3.86 [3.37 to 4.36]
  Shoulder Abduction-Right - Week 9: number analyzed (Participants) | 19 | 19 | 20 | 58
  Shoulder Abduction-Right - Week 9 | -0.19 [-0.95 to 0.56] | 0.22 [-0.50 to 0.95] | 0.12 [-0.28 to 0.51] | 0.05 [-0.30 to 0.40]
  Shoulder Abduction-Right - Week 17: number analyzed (Participants) | 19 | 19 | 19 | 57
  Shoulder Abduction-Right - Week 17 | 0.06 [-0.66 to 0.78] | -0.16 [-1.09 to 0.77] | 0.19 [-0.15 to 0.54] | 0.03 [-0.35 to 0.42]
  Shoulder Abduction-Right - Week 25 | -0.12 [-0.94 to 0.71] | 0.08 [-1.01 to 1.17] | 0.49 [-0.02 to 1.00] | 0.16 [-0.31 to 0.62]
  Shoulder Abduction-Right - Week 33: number analyzed (Participants) | 18 | 19 | 19 | 56
  Shoulder Abduction-Right - Week 33 | -0.16 [-1.26 to 0.94] | -0.54 [-1.32 to 0.24] | 0.42 [0.11 to 0.73] | -0.09 [-0.53 to 0.35]
  Shoulder Abduction-Right - Week 41: number analyzed (Participants) | 19 | 20 | 19 | 58
  Shoulder Abduction-Right - Week 41 | -0.20 [-1.29 to 0.89] | -0.47 [-1.17 to 0.23] | 0.19 [-0.09 to 0.47] | -0.17 [-0.58 to 0.25]
  Shoulder Abduction-Right - Week 49: number analyzed (Participants) | 19 | 20 | 19 | 58
  Shoulder Abduction-Right - Week 49 | 0.35 [-1.48 to 2.18] | -0.43 [-1.02 to 0.16] | 0.66 [0.23 to 1.10] | 0.18 [-0.43 to 0.80]
  Shoulder Abduction-Right - Week 57: number analyzed (Participants) | 18 | 20 | 18 | 56
  Shoulder Abduction-Right - Week 57 | -0.18 [-1.20 to 0.85] | -0.66 [-1.31 to -0.01] | 0.33 [-0.09 to 0.75] | -0.19 [-0.60 to 0.23]
  Shoulder Abduction-Right - Week 65: number analyzed (Participants) | 19 | 20 | 19 | 58
  Shoulder Abduction-Right - Week 65 | -0.10 [-1.10 to 0.90] | -0.16 [-0.98 to 0.67] | 0.25 [-0.08 to 0.57] | -0.01 [-0.43 to 0.42]
  Shoulder Abduction-Right - Week 73 | -0.04 [-1.00 to 0.92] | -0.23 [-0.93 to 0.47] | 0.58 [-0.01 to 1.17] | 0.11 [-0.32 to 0.53]
  Shoulder Abduction-Right - Week 81: number analyzed (Participants) | 19 | 19 | 20 | 58
  Shoulder Abduction-Right - Week 81 | 0.06 [-0.93 to 1.06] | -0.30 [-1.01 to 0.41] | 0.86 [0.26 to 1.46] | 0.22 [-0.22 to 0.66]
  Shoulder Abduction-Right - Week 89: number analyzed (Participants) | 18 | 20 | 19 | 57
  Shoulder Abduction-Right - Week 89 | 0.10 [-0.91 to 1.11] | -0.52 [-1.11 to 0.07] | 0.55 [0.10 to 0.99] | 0.03 [-0.37 to 0.43]
  Shoulder Abduction-Right - Week 97 | -0.02 [-0.96 to 0.92] | -0.28 [-1.08 to 0.53] | 0.46 [-0.27 to 1.19] | 0.06 [-0.40 to 0.51]
  Shoulder Abduction-Right - Week 110: number analyzed (Participants) | 16 | 17 | 17 | 50
  Shoulder Abduction-Right - Week 110 | -0.25 [-1.35 to 0.85] | -0.86 [-1.93 to 0.21] | -0.08 [-0.63 to 0.48] | -0.40 [-0.91 to 0.11]
  Shoulder Abduction-Right - Week 122: number analyzed (Participants) | 11 | 12 | 14 | 37
  Shoulder Abduction-Right - Week 122 | -0.68 [-2.21 to 0.85] | -0.66 [-1.53 to 0.22] | 0.14 [-0.51 to 0.79] | -0.36 [-0.91 to 0.18]
  Shoulder Abduction-Right - Week 146: number analyzed (Participants) | 7 | 6 | 7 | 20
  Shoulder Abduction-Right - Week 146 | -1.50 [-3.96 to 0.96] | -0.75 [-1.89 to 0.39] | 0.19 [-0.44 to 0.81] | -0.69 [-1.52 to 0.15]
  Shoulder Abduction-Right - Week 170: number analyzed (Participants) | 2 | 2 | 2 | 6
  Shoulder Abduction-Right - Week 170 | -4.35 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.90 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -0.20 [NA to NA] — Insufficient number of participants to calculate a 95% Confidence Interval. | -1.82 [-3.95 to 0.31]

49. Secondary Outcome: Serum PF-06252616 (Domagrozumab) Concentration Versus Time Summary
Time Frame: Weeks 1, 25, 49 and 73
Population: The analysis population included all participants who had received at least 1 dose of study medication and had at least 1 PF-06252616 concentration measured in study B5161004. Participants without contributing to the summary statistics are excluded below. Number analyzed refers to number of participants evaluable for specified rows of time points.
Measure: Mean (Standard Deviation); unit: Nanogram Per Milliliter (ng/mL)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3
Number analyzed (Participants) | 14 | 17 | 14
Nanogram Per Milliliter (ng/mL)
  Week 1 | 145774.93 (56594.3925) | 33.3529 (137.5176) | 238433.36 (119862.330)
  Week 25: number analyzed (Participants) | 12 | 12 | 13
  Week 25 | 355111.67 (90842.1052) | 345943.67 (73922.3955) | 488082.31 (199634.909)
  Week 49: number analyzed (Participants) | 7 | 6 | 8
  Week 49 | 405812.43 (110320.246) | 379259.33 (71128.3552) | 459825.13 (49395.4262)
  Week 73: number analyzed (Participants) | 2 | 2 | 2
  Week 73 | 401899.50 (3068.1363) | 400176.00 (84223.4887) | 401847.50 (164854.168)

50. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Development
Description: The criterion for positive result of ADA samples was ADA titer >=1.88. The criterion for negative result of ADA samples was ADA titer <1.88.
Time Frame: Weeks 1, 25, 49, 73 and Early Termination
Population: The analysis population included all participants who had received at least 1 dose of study medication in current study B5161004. Number analyzed refers to the number of participants evaluable for specified rows of time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Participants
  Week 1- Positive >=1.88: number analyzed (Participants) | 14 | 17 | 14 | 45
  Week 1- Positive >=1.88 | 0 | 0 | 0 | 0
  Week 1 - Negative <1.88: number analyzed (Participants) | 14 | 17 | 14 | 45
  Week 1 - Negative <1.88 | 14 | 17 | 14 | 45
  Week 25 - Positive >=1.88: number analyzed (Participants) | 12 | 12 | 13 | 37
  Week 25 - Positive >=1.88 | 0 | 0 | 0 | 0
  Week 25 -Negative <1.88: number analyzed (Participants) | 12 | 12 | 13 | 37
  Week 25 -Negative <1.88 | 12 | 12 | 13 | 37
  Week 49 - Positive >= 1.88: number analyzed (Participants) | 7 | 6 | 8 | 21
  Week 49 - Positive >= 1.88 | 0 | 0 | 0 | 0
  Week 49 -Negative <1.88: number analyzed (Participants) | 7 | 6 | 8 | 21
  Week 49 -Negative <1.88 | 7 | 6 | 8 | 21
  Week 73 - Positive >=1.88: number analyzed (Participants) | 2 | 2 | 2 | 6
  Week 73 - Positive >=1.88 | 0 | 0 | 0 | 0
  Week 73 -Negative <1.88: number analyzed (Participants) | 2 | 2 | 2 | 6
  Week 73 -Negative <1.88 | 2 | 2 | 2 | 6
  Early Termination-Positive>=1.88: number analyzed (Participants) | 17 | 15 | 13 | 45
  Early Termination-Positive>=1.88 | 0 | 0 | 0 | 0
  Early Termination-Negative<1.88: number analyzed (Participants) | 17 | 15 | 13 | 45
  Early Termination-Negative<1.88 | 16 | 14 | 13 | 43

ADVERSE EVENTS:
Time Frame: 2 Years
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Total
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20 | 0/20 | 0/59
Serious Adverse Events (participants affected / at risk) | 2/19 | 2/20 | 1/20 | 5/59
Other Adverse Events (participants affected / at risk) | 15/19 | 17/20 | 17/20 | 49/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sequence 1 (N=19) | Sequence 2 (N=20) | Sequence 3 (N=20) | Total (N=59)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fat embolism syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sequence 1 (N=19) | Sequence 2 (N=20) | Sequence 3 (N=20) | Total (N=59)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (6) | 2 (2) | 3 (3) | 8 (11)
Gait inability (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (5) | 2 (5)
Pyrexia (General disorders) | 2 (3) | 3 (3) | 1 (1) | 6 (7)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 5 (5)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3) | 4 (5) | 11 (12)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1/16 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 2 (2) | 5 (6)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 3 (5) | 6 (12) | 13 (22)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insulin resistance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 5 (8) | 1 (1) | 5 (12) | 11 (21)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (4) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 6 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 3 (4) | 5 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to insufficient efficacy and not due to safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT02907619/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT02907619/SAP_001.pdf